CLINICAL TRIAL: NCT02608268
Title: Phase I-Ib/II Open-label Multi-center Study of the Safety and Efficacy of MBG453 as Single Agent and in Combination With PDR001 in Adult Patients With Advanced Malignancies
Brief Title: Phase I-Ib/II Study of MBG453 as Single Agent and in Combination With PDR001 in Patients With Advanced Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMBG453X2101; 2015-002354-12 (EudraCT Number)
Record Dates: First submitted 2015-10-15; First posted 2015-11-18 (Estimated); Results first posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Advanced Malignancies
Keywords: Solid tumors; Melanoma; Non small cell lung cancer; NSCLC; Renal cell carcinoma; RCC; Phase I-Ib/II; MBG453; PDR001; Checkpoint inhibitor; PD-1; TIM-3
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell | interventions — sabatolimab; spartalizumab; Decitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Phase I Dose escalation: MBG453 Q2W ROW (Experimental): Sabatolimab every 2 weeks (Q2W) in Phase I Dose Escalation Part in rest of the world (ROW) patients
  Interventions: Drug: MBG453
- Phase I Dose escalation: MBG453 Q2W Japan (Experimental): Sabatolimab Q2W in Phase I Dose Escalation Part in Japanese patients
  Interventions: Drug: MBG453
- Phase I Dose escalation: MBG453 Q4W ROW (Experimental): Sabatolimab every 4 weeks (Q4W) in Phase I Dose Escalation Part in ROW patients
  Interventions: Drug: MBG453
- Phase I Dose escalation: MBG453 Q4W Japan (Experimental): Sabatolimab Q4W in Phase I Dose Escalation Part in Japanese patients
  Interventions: Drug: MBG453
- Phase Ib Dose Escalation: MBG453 Q2W + PDR001 Q2W (Experimental): Sabatolimab Q2W in combination with spartalizumab Q2W in Phase Ib Dose Escalation Part
  Interventions: Drug: MBG453; Drug: PDR001
- Phase Ib Dose Escalation: MBG453 Q4W + PDR001 Q4W (Experimental): Sabatolimab Q4W in combination with spartalizumab Q4W in Phase Ib Dose Escalation Part
  Interventions: Drug: MBG453; Drug: PDR001
- Phase Ib Dose Escalation: MBG453 + Decitabine (Experimental): Sabatolimab in combination with decitabine in Phase Ib Dose Escalation Part. This arm was not opened for enrollment.
  Interventions: Drug: MBG453; Drug: Decitabine
- Dose Ranging Part: MBG453 Q4W (Experimental): Sabatolimab Q4W in Dose Ranging Part
  Interventions: Drug: MBG453
- Phase II: MBG453 + PDR001 (Experimental): Sabatolimab Q4W in combination with spartalizumab Q4W in non-small cell lung carcinoma (NSCLC) and melanoma
  Interventions: Drug: MBG453; Drug: PDR001
- Phase II: MBG453 (Experimental): Sabatolimab alone in Phase II. This arm was not opened for enrollment.
  Interventions: Drug: MBG453

INTERVENTIONS:
Drug: MBG453 — Anti human TIM-3 monoclonal antibody. MBG453 administered via intravenous (i.v.) infusion either every 2 weeks (Q2W) or every 4 weeks (Q4W).
  Other Names: sabatolimab
Drug: PDR001 — Anti-human PD-1 monoclonal antibody. PDR001 administered via intravenous (i.v.) infusion either every 2 weeks (Q2W) or every 4 weeks (Q4W).
  Other Names: spartalizumab
  Arms: Phase II: MBG453 + PDR001; Phase Ib Dose Escalation: MBG453 Q2W + PDR001 Q2W; Phase Ib Dose Escalation: MBG453 Q4W + PDR001 Q4W
Drug: Decitabine — commercially available chemotherapy
  Arms: Phase Ib Dose Escalation: MBG453 + Decitabine

SUMMARY:
The purpose of this first-in-human study of MBG453 was to characterize the safety, tolerability, pharmacokinetics, pharmacodynamics and anti-tumor activity of MBG453 administered i.v. as a single agent or in combination with PDR001 or decitabine in adult patients with advanced solid tumors

DETAILED DESCRIPTION:
This study was a first in human (FIH), open-label, Phase I-Ib/II, multi-center study which consisted of a Phase I dose escalation part of sabatolimab (MBG453) as single agent, and a Phase Ib dose escalation part of sabatolimab in combination with spartalizumab (PDR001) that commenced after two cohorts in the dose escalation with single agent were completed. Once the maximum tolerated dose (MTD)/recommended Phase II dose (RP2D) of sabatolimab as single agent and in combination with spartalizumab was achieved, a dose ranging part and a Phase II part started.

• Phase I dose escalation part (sabatolimab single agent): In the Phase I part of the study, cohorts of subjects were treated with sabatolimab as single agent either every 2 weeks (Q2W) or every 4 weeks (Q4W) until the MTD was reached or a lower RP2D was established.

The sabatolimab single agent dose escalation part in Japan ran separately in order to ensure that the safety and pharmacokinetics (PK) profiles of single-agent sabatolimab are adequately characterized in Japanese patients. If the recommended dose of single agent sabatolimab in Japanese patients was the same as in the rest of the world (ROW) patients, then patients enrolled in Japan were to be recruited into the other parts of the study.

• Phase Ib dose escalation part (sabatolimab in combination with spartalizumab): The combination Phase Ib part of the study was to be commenced after at least two cohorts of sabatolimab as single agent were completed, and safety data suggested acceptable toxicity for subjects to begin treatment in combination. Following identification of the MTD/RP2D for the combination of sabatolimab and spartalizumab with a Q2W dosing schedule, a further dose escalation was planned to identify the MTD/RP2D with a Q4W dosing schedule.

The sabatolimab in combination with decitabine treatment arm (Phase Ib) was not opened for enrollment.

* Dose ranging part: During the dose ranging part various dose levels of single agent sabatolimab were tested to better understand the safety, tolerability and PK.
* Phase II part (sabatolimab in combination with spartalizumab): Once the MTD and/or RP2D were declared for sabatolimab in combination with spartalizumab, additional subjects were enrolled in the Phase II part in the selected indications (melanoma and non-small cell lung carcinoma) in order to assess the preliminary anti-tumor activity.

The Phase II single agent sabatolimab treatment arm was not opened for enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented advanced or metastatic solid tumors.
* Phase I-Ib part (including dose ranging part): Patients with advanced/metastatic solid tumors, with measurable or non-measurable disease as determined by RECIST v1.1, who have progressed despite standard therapy or are intolerant of standard therapy, or for whom no standard therapy exists and who did not receive prior anti-PD-1/PD-L1 treatment.
* Phase II part (MBG453 single agent): Patients with advanced/metastatic solid tumors in the indication in which at least one confirmed PR or CR was seen during the dose escalation phase I part. Patients must have measurable disease as determined by RECIST v1.1, have progressed despite standard therapy or be intolerant to standard therapy.
* Phase II part (MBG453 in combination PDR001): Patients with advanced/metastatic tumors in the below selected indications, with at least one measurable lesion as determined by RECIST v1.1, who have received standard therapy and are intolerant of standard therapy or have progressed following their last prior therapy.:

  * Melanoma (anti-PD-1/PD-L1 therapy naïve or pre-treated)
  * Non small cell lung cancer (anti-PD-1/PD-L1 therapy naïve or pre-treated)
  * Renal Cell Carcinoma (anti-PD-1/PD-L1 therapy naïve or pre-treated)
* Must have a site of disease amenable to biopsy, and be a candidate for tumor biopsy according to the treating institution's guidelines. Patient must be willing to undergo a new tumor biopsy at screening/baseline, and during therapy on the study.
* For MBG453 in combination with decitabine: anti-PD-1/PD-L1 therapy naïve SCLC patients who have failed no more than two lines of standard chemotherapy including topotecan

Exclusion Criteria:

* Presence of symptomatic central nervous system metastases.
* History of severe hypersensitivity reactions to other monoclonal antibodies.
* Human Immunodeficiency Virus, Hepatitis B Virus or Hepatitis C Virus infection.
* Active autoimmune disease or a documented history of autoimmune disease, including ulcerative colitis and Crohn's disease or any condition that requires systemic steroids.
* Systemic steroid therapy or any immunosuppressive therapy (≥10mg/day prednisone or equivalent).
* Use of any vaccines against infectious diseases (e.g. varicella, pneumococcus) within 4 weeks of initiation of study treatment.
* Pre-treatment with anti-CTLA4 antibodies in combination with any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathway.
* Participation in an interventional, investigational non-immunotherapy study within 2 weeks of the first dose of study treatment.
* Prior participation in an interventional, investigational cancer vaccine or immunotherapy study except for an anti-PD-1/PD-L1 study.
* For MBG453 in combination with decitabine: Hypersensitivity to decitabine or to any of the excipients, listed in decitabine country specific label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2015-11-23 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (14):
- United States (4):
  - Sidney Kimmel CCC At JH Sidney Kimmel CCC, Baltimore, Maryland
  - Dana Farber Cancer Institute DFCI - Brookline, Boston, Massachusetts
  - UT M.D Anderson Cancer Center, Houston, Texas
  - Mays Cancer Ctr Uthsa Mdacc, San Antonio, Texas
- Novartis Investigative Site, Toronto, Ontario, Canada
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
- Novartis Investigative Site, Kashiwa, Chiba, Japan
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Leiden
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Novartis Investigative Site, Geneva, Switzerland
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Lin CC, Curigliano G, Santoro A, Kim DW, Tai D, Hodi FS, Wilgenhof S, Doi T, Sabatos-Peyton C, Szpakowski S, Chitnis S, Xyrafas A, Gutzwiller S, Pastore A, Mach N. Sabatolimab in combination with spartalizumab in patients with non-small cell lung cancer or melanoma who received prior treatment with anti-PD-1/PD-L1 therapy: a phase 2 multicentre study. BMJ Open. 2024 Aug 29;14(8):e079132. doi: 10.1136/bmjopen-2023-079132. PMID 39209782
- [Derived] Curigliano G, Gelderblom H, Mach N, Doi T, Tai D, Forde PM, Sarantopoulos J, Bedard PL, Lin CC, Hodi FS, Wilgenhof S, Santoro A, Sabatos-Peyton CA, Longmire TA, Xyrafas A, Sun H, Gutzwiller S, Manenti L, Naing A. Phase I/Ib Clinical Trial of Sabatolimab, an Anti-TIM-3 Antibody, Alone and in Combination with Spartalizumab, an Anti-PD-1 Antibody, in Advanced Solid Tumors. Clin Cancer Res. 2021 Jul 1;27(13):3620-3629. doi: 10.1158/1078-0432.CCR-20-4746. Epub 2021 Apr 21. PMID 33883177

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 14 investigative sites in 9 countries.
Pre-assignment Details: The screening period began once patients had signed the study informed consent. Screening evaluations were performed within 28 days prior to the first dose of study medication. After screening, the treatment period started on Cycle 1 Day 1.
Groups:
- Phase I Dose Escalation: MBG453 80mg Q2W ROW: Sabatolimab 80 mg every 2 weeks (Q2W) in Phase I Dose Escalation Part in rest of the world (ROW) patients
- Phase I Dose Escalation: MBG453 240mg Q2W ROW: Sabatolimab 240 mg Q2W in Phase I Dose Escalation Part in ROW patients
- Phase I Dose Escalation: MBG453 800mg Q2W ROW: Sabatolimab 800 mg Q2W in Phase I Dose Escalation Part in ROW patients
- Phase I Dose Escalation: MBG453 1200mg Q2W ROW: Sabatolimab 1200 mg Q2W in Phase I Dose Escalation Part in ROW patients
- Phase I Dose Escalation: MBG453 80mg Q2W Japan: Sabatolimab 80 mg Q2W in Phase I Dose Escalation Part in Japanese patients
- Phase I Dose Escalation: MBG453 240mg Q2W Japan: Sabatolimab 240 mg Q2W in Phase I Dose Escalation Part in Japanese patients
- Phase I Dose Escalation: MBG453 800mg Q2W Japan: Sabatolimab 800 mg Q2W in Phase I Dose Escalation Part in Japanese patients
- Phase I Dose Escalation: MBG453 1200mg Q2W Japan: Sabatolimab 1200 mg Q2W in Phase I Dose Escalation Part in Japanese participants
- Phase I Dose Escalation: MBG453 240mg Q4W ROW: Sabatolimab 240 mg every 4 weeks (Q4W) in Phase I Dose Escalation Part in ROW patients
- Phase I Dose Escalation: MBG453 800mg Q4W ROW: Sabatolimab 800 mg Q4W in Phase I Dose Escalation Part in ROW patients
- Phase I Dose Escalation: MBG453 1200mg Q4W ROW: Sabatolimab 1200 mg Q4W in Phase I Dose Escalation Part in ROW patients
- Phase I Dose Escalation: MBG453 1200mg Q4W Japan: Sabatolimab 1200 mg Q4W in Phase I Dose Escalation Part in Japanese patients
- Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W: Sabatolimab 20 mg Q2W in combination with spartalizumab 80 mg Q2W in Phase Ib Dose Escalation Part
- Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W: Sabatolimab 80 mg Q2W in combination with spartalizumab 80 mg Q2W in Phase Ib Dose Escalation Part
- Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W: Sabatolimab 240 mg Q2W in combination with spartalizumab 80 mg Q2W in Phase Ib Dose Escalation Part
- Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W: Sabatolimab 240 mg Q2W in combination with spartalizumab 240 mg Q2W in Phase Ib Dose Escalation Part
- Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W: Sabatolimab 800 mg Q2W in combination with spartalizumab 80 mg Q2W in Phase Ib Dose Escalation Part
- Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W: Sabatolimab 800 mg Q2W in combination with spartalizumab 240 mg Q2W in Phase Ib Dose Escalation Part
- Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W: Sabatolimab 80 mg Q4W in combination with spartalizumab 80 mg Q4W in Phase Ib Dose Escalation Part
- Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W: Sabatolimab 80 mg Q4W in combination with spartalizumab 400 mg Q4W in Phase Ib Dose Escalation Part
- Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W: Sabatolimab 240 mg Q4W in combination with spartalizumab 80 mg Q4W in Phase Ib Dose Escalation Part
- Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W: Sabatolimab 240 mg Q4W in combination with spartalizumab 240 mg Q4W in Phase Ib Dose Escalation Part
- Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W: Sabatolimab 240 mg Q4W in combination with spartalizumab 400 mg Q4W in Phase Ib Dose Escalation Part
- Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W: Sabatolimab 800 mg Q4W in combination with spartalizumab 400 mg Q4W in Phase Ib Dose Escalation Part
- Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W: Sabatolimab 1200 mg Q4W in combination with spartalizumab 400 mg Q4W in Phase Ib Dose Escalation Part
- Dose Ranging Part: MBG453 80mg Q4W: Sabatolimab 80 mg Q4W in Dose Ranging Part
- Dose Ranging Part: MBG453 240mg Q4W: Sabatolimab 240 mg Q4W in Dose Ranging Part
- Dose Ranging Part: MBG453 1200mg Q4W: Sabatolimab 1200 mg Q4W in Dose Ranging Part
- Phase II: MBG453 + PDR001 NSCLC: Sabatolimab 800 mg Q4W in combination with spartalizumab 400 mg Q4W in non-small cell lung carcinoma (NSCLC)
- Phase II: MBG453 + PDR001 Melanoma: Sabatolimab 800 mg Q4W in combination with spartalizumab 400 mg Q4W in melanoma
Period: Overall Study
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Started | 14 | 9 | 16 | 5 | 2 | 4 | 6 | 2 | 8 | 9 | 6 | 6 | 6 | 13 | 6 | 5 | 5 | 6 | 6 | 3 | 12 | 5 | 7 | 6 | 6 | 14 | 17 | 15 | 17 | 16
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 14 | 9 | 16 | 5 | 2 | 4 | 6 | 2 | 8 | 9 | 6 | 6 | 6 | 13 | 6 | 5 | 5 | 6 | 6 | 3 | 12 | 5 | 7 | 6 | 6 | 14 | 17 | 15 | 17 | 16
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 4 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 1
Not completed — Progressive disease | 12 | 8 | 13 | 5 | 2 | 4 | 6 | 2 | 5 | 6 | 5 | 5 | 4 | 11 | 6 | 3 | 5 | 5 | 5 | 2 | 10 | 4 | 5 | 5 | 3 | 11 | 16 | 11 | 10 | 15
Not completed — Subject/guardian decision | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma | Total
Number analyzed (Participants) | 14 | 9 | 16 | 5 | 2 | 4 | 6 | 2 | 8 | 9 | 6 | 6 | 6 | 13 | 6 | 5 | 5 | 6 | 6 | 3 | 12 | 5 | 7 | 6 | 6 | 14 | 17 | 15 | 17 | 16 | 252
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (13.80) | 50.7 (16.69) | 53.6 (15.95) | 57.2 (8.07) | 73.0 (8.49) | 65.8 (5.74) | 54.0 (16.64) | 55.0 (7.07) | 56.1 (12.76) | 62.2 (10.86) | 60.8 (13.09) | 63.5 (7.40) | 47.8 (13.92) | 56.9 (13.98) | 56.5 (16.56) | 54.6 (15.87) | 56.0 (10.58) | 54.0 (12.77) | 54.2 (14.47) | 62.3 (22.37) | 66.0 (7.02) | 59.4 (20.16) | 61.3 (14.51) | 53.8 (10.36) | 57.7 (12.16) | 57.4 (12.20) | 59.4 (10.12) | 57.3 (11.85) | 64.5 (10.28) | 61.8 (11.35) | 58.4 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 5 | 3 | 1 | 2 | 4 | 1 | 6 | 4 | 3 | 3 | 2 | 7 | 2 | 2 | 0 | 4 | 3 | 2 | 5 | 2 | 3 | 4 | 3 | 10 | 14 | 13 | 3 | 8 | 132
  Male | 6 | 4 | 11 | 2 | 1 | 2 | 2 | 1 | 2 | 5 | 3 | 3 | 4 | 6 | 4 | 3 | 5 | 2 | 3 | 1 | 7 | 3 | 4 | 2 | 3 | 4 | 3 | 2 | 14 | 8 | 120
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 12 | 9 | 12 | 4 | 0 | 0 | 0 | 0 | 7 | 9 | 5 | 0 | 2 | 11 | 4 | 4 | 2 | 4 | 3 | 2 | 10 | 4 | 5 | 3 | 5 | 12 | 15 | 14 | 11 | 8 | 177
  Asian | 1 | 0 | 3 | 1 | 2 | 4 | 6 | 2 | 1 | 0 | 1 | 6 | 3 | 2 | 2 | 1 | 3 | 1 | 3 | 1 | 2 | 1 | 2 | 2 | 1 | 1 | 1 | 0 | 5 | 8 | 66
  Black | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 4
  Unknown | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Other | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Phase I-Ib and Dose Ranging Part: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) During the On-treatment Period
Description: Number of participants with AEs (any AE regardless of seriousness) and SAEs, including changes from baseline in vital signs, electrocardiograms and laboratory results qualifying and reported as AEs.
  AE grades to characterize the severity of the AEs were based on the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. For CTCAE v4.03, Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = death related to AE.
  The on-treatment period is defined from the day of first administration of study treatment up to 30 days after the date of its last administration.
Time Frame: From first dose of study medication up to 30 days after last dose, with a maximum duration of 2 years for sabatolimab and 5 years for sabatolimab in combination with spartalizumab
Population: All patients in Phase I-Ib and Dose ranging Part who received at least one dose of assigned single agent sabatolimab, or at least one full or partial dose of assigned combination sabatolimab+spartalizumab
Measure: Count of Participants; unit: Participants
Groups:
- Phase I Dose Escalation: MBG453 80mg Q2W ROW: Sabatolimab 80 mg Q2W in Phase I Dose Escalation Part in ROW patients
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W
Number analyzed (Participants) | 14 | 9 | 16 | 5 | 2 | 4 | 6 | 2 | 8 | 9 | 6 | 6 | 6 | 13 | 6 | 5 | 5 | 6 | 6 | 3 | 12 | 5 | 7 | 6 | 6 | 14 | 17 | 15
Participants
  AEs | 13 | 9 | 14 | 5 | 2 | 3 | 6 | 2 | 7 | 9 | 6 | 5 | 6 | 12 | 6 | 5 | 5 | 6 | 6 | 3 | 11 | 5 | 7 | 6 | 6 | 13 | 17 | 14
  Treatment-related AEs | 9 | 5 | 6 | 1 | 0 | 0 | 1 | 0 | 4 | 6 | 2 | 1 | 5 | 7 | 5 | 4 | 2 | 4 | 3 | 1 | 5 | 5 | 3 | 4 | 2 | 3 | 7 | 10
  AEs with grade ≥ 3 | 5 | 3 | 6 | 2 | 0 | 1 | 2 | 0 | 3 | 7 | 4 | 3 | 4 | 9 | 3 | 5 | 3 | 0 | 4 | 1 | 3 | 3 | 6 | 5 | 4 | 10 | 7 | 10
  Treatment-related AEs with grade ≥ 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 2
  SAEs | 4 | 1 | 6 | 2 | 0 | 0 | 0 | 0 | 1 | 5 | 4 | 0 | 2 | 6 | 2 | 4 | 4 | 0 | 4 | 1 | 2 | 3 | 1 | 3 | 3 | 8 | 7 | 7
  Fatal SAEs | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  AEs leading to discontinuation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0
  AEs leading to dose adjustment/interruption | 3 | 0 | 3 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 1 | 3 | 3 | 3 | 1 | 3 | 1 | 1 | 1 | 1 | 0 | 1 | 2 | 2 | 1 | 0 | 2
  AEs requiring additional therapy | 13 | 4 | 12 | 4 | 2 | 3 | 6 | 2 | 7 | 7 | 3 | 3 | 5 | 12 | 4 | 5 | 4 | 4 | 6 | 3 | 10 | 5 | 3 | 6 | 5 | 12 | 17 | 12

2. Primary Outcome: Phase I-Ib: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value of Common Terminology Criteria for Adverse Events (CTCAE) grade ≥ 3 assessed as unrelated to disease, disease progression, inter-current illness or concomitant medications, which occurs within the first cycle of treatment with sabatolimab as single agent or in the first two cycles of treatment when sabatolimab is given in combination with spartalizumab during the dose escalation part of the study. Other clinically significant toxicities may be considered to be DLTs, even if not CTCAE grade 3 or higher. The duration of one treatment cycle is 28 days.
Time Frame: 28 days (sabatolimab single agent) and 56 days (sabatolimab+spartalizumab)
Population: Patients in Phase I-Ib who either met the minimum exposure criterion defined in the protocol and had sufficient safety evaluations, or had experienced a DLT during Cycle 1 or Cycle 2 (combination arm only)
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W
Number analyzed (Participants) | 13 | 9 | 12 | 5 | 2 | 4 | 6 | 2 | 8 | 8 | 5 | 6 | 6 | 12 | 4 | 4 | 5 | 5 | 6 | 2 | 12 | 5 | 5 | 4 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

3. Primary Outcome: Phase I-Ib and Dose Ranging Part: Number of Participants With Dose Reductions and Dose Interruptions of Sabatolimab
Description: Number of participants with at least one dose reduction of sabatolimab and number of participants with at least one dose interruption of sabatolimab.
Time Frame: From first dose of study medication up to last dose, with a maximum duration of 1.9 years for sabatolimab and 4.9 years for sabatolimab in combination with spartalizumab
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W
Number analyzed (Participants) | 14 | 9 | 16 | 5 | 2 | 4 | 6 | 2 | 8 | 9 | 6 | 6 | 6 | 13 | 6 | 5 | 5 | 6 | 6 | 3 | 12 | 5 | 7 | 6 | 6 | 14 | 17 | 15
Participants
  At least one dose reduction | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  At least one dose interruption | 2 | 1 | 3 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 1

4. Primary Outcome: Phase Ib: Number of Participants With Dose Reductions and Dose Interruptions of Spartalizumab
Description: Number of participants with at least one dose reduction of spartalizumab and number of participants with at least one dose interruption of spartalizumab.
Time Frame: From first dose of study medication up to last dose, with a maximum duration of 4.9 years
Population: All patients in Phase Ib who received at least one full or partial dose of assigned combination sabatolimab+spartalizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W
Number analyzed (Participants) | 6 | 13 | 6 | 5 | 5 | 6 | 6 | 3 | 12 | 5 | 7 | 6 | 6
Participants
  At least one dose reduction | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  At least one dose interruption | 2 | 2 | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 1

5. Primary Outcome: Phase I-Ib and Dose Ranging Part: Dose Intensity of Sabatolimab
Description: Dose intensity of sabatolimab Q2W was calculated as cumulative actual dose in milligrams divided by duration of exposure in days and then multiplied by 14 days.
  Dose intensity of sabatolimab Q4W was calculated as cumulative actual dose in milligrams divided by duration of exposure in days and then multiplied by 28 days.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W
Number analyzed (Participants) | 14 | 9 | 16 | 5 | 2 | 4 | 6 | 2 | 8 | 9 | 6 | 6 | 6 | 13 | 6 | 5 | 5 | 6 | 6 | 3 | 12 | 5 | 7 | 6 | 6 | 14 | 17 | 15
milligrams | 78.35 (4.678) | 235.60 (17.140) | 728.06 (164.525) | 1203.03 (15.891) | 80.00 (0.000) | 217.50 (28.723) | 758.03 (57.03) | 1208.70 (12.298) | 240.19 (1.954) | 752.29 (123.021) | 1193.10 (16.893) | 1196.49 (8.595) | 19.34 (1.043) | 78.58 (2.872) | 236.19 (15.050) | 230.24 (19.982) | 743.88 (79.534) | 763.72 (89.571) | 76.39 (5.315) | 80.11 (0.184) | 239.36 (4.227) | 236.00 (7.800) | 230.28 (21.179) | 755.79 (103.897) | 1196.15 (9.421) | 79.55 (1.661) | 239.68 (4.977) | 1192.33 (23.366)

6. Primary Outcome: Phase Ib: Dose Intensity of Spartalizumab
Description: Dose intensity of spartalizumab Q2W was calculated as cumulative actual dose in milligrams divided by duration of exposure in days and then multiplied by 14 days.
  Dose intensity of spartalizumab Q4W was calculated as cumulative actual dose in milligrams divided by duration of exposure in days and then multiplied by 28 days.
Time Frame: From first dose of study medication up to last dose, with a maximum duration of 4.9 years
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W
Number analyzed (Participants) | 6 | 13 | 6 | 5 | 5 | 6 | 6 | 3 | 12 | 5 | 7 | 6 | 6
milligrams | 77.36 (4.171) | 77.83 (3.957) | 78.73 (5.017) | 230.24 (19.982) | 74.39 (7.953) | 229.12 (26.871) | 76.39 (5.315) | 400.53 (0.920) | 79.79 (1.409) | 236.00 (7.800) | 383.22 (36.754) | 377.89 (51.948) | 398.72 (3.140)

7. Primary Outcome: Phase II: Overall Response Rate (ORR) Per RECIST v1.1
Description: Tumor response was based on local investigator assessment as per Response Evaluation Criteria In Solid Tumors (RECIST) v1.1. ORR per RECIST v1.1 is defined as the percentage of participants with a best overall response of Complete Response (CR) or Partial Response (PR).
  For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: From start of treatment until end of treatment, assessed up to 2.9 years
Population: All patients in Phase II who received at least one full or partial dose of the combination sabatolimab+spartalizumab
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 17 | 16
Percentage of participants | 0 [0.0 to 16.2] | 0 [0.0 to 17.1]

8. Secondary Outcome: Best Overall Response (BOR) Per RECIST v1.1
Description: BOR is defined as the best response recorded from the start of the study treatment until disease progression/recurrence, based on local investigator assessment per RECIST v1.1.
  For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters; PD= At least a 20% increase in the sum of diameters of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition, the sum must also demonstrate an absolute increase of at least 5 mm; SD= Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progression; NCRNPD: Persistence of one or more non-target lesions.
  Number of participants in each category is reported in the table.
Time Frame: From start of treatment until end of treatment, assessed up to 1.9 years for sabatolimab and 4.9 years for sabatolimab in combination with spartalizumab
Population: All patients who received at least one dose of assigned single agent sabatolimab, or at least one full or partial dose of assigned combination sabatolimab+spartalizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 14 | 9 | 16 | 5 | 2 | 4 | 6 | 2 | 8 | 9 | 6 | 6 | 6 | 13 | 6 | 5 | 5 | 6 | 6 | 3 | 12 | 5 | 7 | 6 | 6 | 14 | 17 | 15 | 17 | 16
Participants
  Complete Response (CR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response (PR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Stable Disease (SD) | 4 | 3 | 7 | 0 | 0 | 1 | 2 | 0 | 3 | 1 | 0 | 3 | 4 | 7 | 2 | 1 | 1 | 1 | 3 | 1 | 5 | 3 | 2 | 2 | 1 | 4 | 2 | 4 | 6 | 3
  Progressive Disease (PD) | 7 | 6 | 8 | 5 | 2 | 3 | 4 | 2 | 3 | 4 | 4 | 3 | 1 | 4 | 4 | 4 | 3 | 4 | 3 | 1 | 7 | 2 | 1 | 3 | 3 | 7 | 13 | 8 | 5 | 12
  Non-CR/Non-PD (NCRNPD) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 3 | 2 | 3 | 6 | 1

9. Secondary Outcome: Progression-Free Survival (PFS) Per RECIST v1.1
Description: PFS is defined as the time from the date of start of treatment to the date of the first documented progression or death due to any cause. If a patient did not have an event, PFS was censored at the date of the last adequate tumor assessment. Tumor response was based on local investigator assessment per RECIST v1.1.
  PFS was analyzed using Kaplan-Meier estimates.
Time Frame: From start of treatment until first documented progression or death due to any cause, assessed up to 1.9 years for sabatolimab and 4.9 years for sabatolimab in combination with spartalizumab
Population: as for outcome 8
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 14 | 9 | 16 | 5 | 2 | 4 | 6 | 2 | 8 | 9 | 6 | 6 | 6 | 13 | 6 | 5 | 5 | 6 | 6 | 3 | 12 | 5 | 7 | 6 | 6 | 14 | 17 | 15 | 17 | 16
months | 1.8 [1.7 to 3.3] | 1.8 [1.6 to 2.8] | 1.8 [1.7 to 5.3] | 1.7 [1.3 to NA] — Not estimable due to insufficient number of participants with events. | 1.5 [1.4 to NA] — Not estimable due to insufficient number of participants with events. | 1.9 [1.0 to NA] — Not estimable due to insufficient number of participants with events. | 2.0 [1.0 to 3.3] | 1.6 [1.4 to NA] — Not estimable due to insufficient number of participants with events. | 1.7 [1.0 to NA] — Not estimable due to insufficient number of participants with events. | 1.7 [0.7 to 1.8] | 1.8 [1.6 to NA] — Not estimable due to insufficient number of participants with events. | 2.0 [1.1 to 3.5] | 3.6 [1.8 to NA] — Not estimable due to insufficient number of participants with events. | 3.6 [1.8 to 3.7] | 1.7 [1.0 to 3.7] | 1.8 [1.0 to NA] — Not estimable due to insufficient number of participants with events. | 1.8 [1.7 to NA] — Not estimable due to insufficient number of participants with events. | 1.7 [0.5 to 1.8] | 2.6 [1.6 to 3.7] | 2.4 [1.8 to NA] — Not estimable due to insufficient number of participants with events. | 1.8 [1.7 to 3.0] | 3.5 [1.8 to NA] — Not estimable due to insufficient number of participants with events. | NA [1.5 to NA] — Not estimable due to insufficient number of participants with events. | 2.7 [1.1 to 3.8] | 1.7 [0.2 to 2.4] | 1.8 [1.7 to 3.7] | 1.7 [1.6 to 1.8] | 1.7 [1.7 to 2.1] | 1.7 [1.1 to 3.4] | 1.8 [1.7 to 1.9]

10. Secondary Outcome: Duration of Response (DOR) Per RECIST v1.1
Description: DOR only applies to patients for whom best overall response is complete response (CR) or partial response (PR) based on local investigator assessment according to RECIST v1.1. DOR is defined as the time from the date of first documented response to the date of first documented progression or death due to underlying cancer. If a patient did not have an event, duration was censored at the date of last adequate tumor assessment.
  According to the statistical analysis plan (SAP), summary estimates of DOR using the Kaplan-Meier method were planned to be reported if there were at least 10 patients achieving a confirmed CR or PR in each treatment group/arm.
Time Frame: From first documented response to first documented disease progression or death due to underlying cancer, assessed up to 1.9 years for sabatolimab and 4.9 years for sabatolimab in combination with spartalizumab
Population: All patients for whom best overall response is complete response (CR) or partial response (PR) per RECIST v1.1
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
months |  |  |  |  |  |  |  |  |  |  |  |  | NA [NA to NA] — The estimate could not be provided due to the insufficient number of responders as per SAP. | NA [NA to NA] — The estimate could not be provided due to the insufficient number of responders as per SAP. |  |  |  |  |  |  |  |  | NA [NA to NA] — The estimate could not be provided due to the insufficient number of responders as per SAP. | NA [NA to NA] — The estimate could not be provided due to the insufficient number of responders as per SAP. |  |  |  |  |  |

11. Secondary Outcome: Overall Response Rate (ORR) Per irRC
Description: Tumor response was based on local investigator assessment as per irRC. ORR per irRC is defined as the percentage of participants with a best overall response of immune related Complete Response (irCR) or immune related Partial Response (irPR).
  For irRC, irCR=Disappearance of all non-nodal target lesions and non-target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; irPR= At least a 30% decrease in the sum of diameters of all target lesions including new measurable lesions, taking as reference the baseline sum of diameters.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 14 | 9 | 16 | 5 | 2 | 4 | 6 | 2 | 8 | 9 | 6 | 6 | 6 | 13 | 6 | 5 | 5 | 6 | 6 | 3 | 12 | 5 | 7 | 6 | 6 | 14 | 17 | 15 | 17 | 16
Percentage of participants | 0 [0.0 to 19.3] | 0 [0.0 to 28.3] | 0 [0.0 to 17.1] | 0 [0.0 to 45.1] | 0 [0.0 to 77.6] | 0 [0.0 to 52.7] | 0 [0.0 to 39.3] | 0 [0.0 to 77.6] | 0 [0.0 to 31.2] | 0 [0.0 to 28.3] | 0 [0.0 to 39.3] | 0 [0.0 to 39.3] | 16.7 [0.9 to 58.2] | 7.7 [0.4 to 31.6] | 0 [0.0 to 39.3] | 0 [0.0 to 45.1] | 0 [0.0 to 45.1] | 0 [0.0 to 39.3] | 0 [0.0 to 39.3] | 0 [0.0 to 63.2] | 0 [0.0 to 22.1] | 0 [0.0 to 45.1] | 28.6 [5.3 to 65.9] | 16.7 [0.9 to 58.2] | 0 [0.0 to 39.3] | 0 [0.0 to 19.3] | 0 [0.0 to 16.2] | 0 [0.0 to 18.1] | 0 [0.0 to 16.2] | 0 [0.0 to 17.1]

12. Secondary Outcome: Progression-Free Survival (PFS) Per irRC
Description: PFS is defined as the time from the date of start of treatment to the date of the first documented and confirmed progression or death due to any cause. If a patient did not have an event, PFS was censored at the date of the last adequate tumor evaluation. Tumor response was based on local investigator assessment per irRC.
  PFS was analyzed using Kaplan-Meier estimates.
Time Frame: From start of treatment until first documented and confirmed progression or death due to any cause, assessed up to 1.9 years for sabatolimab and 4.9 years for sabatolimab in combination with spartalizumab
Population: as for outcome 8
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 14 | 9 | 16 | 5 | 2 | 4 | 6 | 2 | 8 | 9 | 6 | 6 | 6 | 13 | 6 | 5 | 5 | 6 | 6 | 3 | 12 | 5 | 7 | 6 | 6 | 14 | 17 | 15 | 17 | 16
months | 1.8 [1.7 to 3.3] | 1.8 [1.6 to 3.0] | 1.8 [1.7 to 5.3] | 1.7 [1.3 to NA] — Not estimable due to insufficient number of participants with events. | 1.5 [1.4 to NA] — Not estimable due to insufficient number of participants with events. | 1.9 [1.0 to NA] — Not estimable due to insufficient number of participants with events. | 2.0 [1.0 to 3.3] | 1.6 [1.4 to NA] — Not estimable due to insufficient number of participants with events. | 1.7 [1.0 to NA] — Not estimable due to insufficient number of participants with events. | 1.8 [0.7 to 2.5] | 2.3 [1.8 to NA] — Not estimable due to insufficient number of participants with events. | 2.0 [1.1 to 3.5] | 3.6 [1.8 to NA] — Not estimable due to insufficient number of participants with events. | 3.6 [1.8 to 3.7] | 1.7 [1.0 to 3.7] | 1.8 [1.0 to NA] — Not estimable due to insufficient number of participants with events. | 1.8 [1.7 to NA] — Not estimable due to insufficient number of participants with events. | 1.7 [0.5 to 1.8] | 2.6 [1.6 to 3.7] | 2.4 [1.8 to NA] — Not estimable due to insufficient number of participants with events. | 2.3 [1.7 to 3.6] | 5.5 [3.5 to NA] — Not estimable due to insufficient number of participants with events. | NA [1.5 to NA] — Not estimable due to insufficient number of participants with events. | 2.7 [1.1 to 3.8] | 1.7 [0.2 to 2.4] | 1.8 [1.7 to 3.2] | 1.7 [1.6 to 1.8] | 1.7 [1.7 to 2.1] | 1.7 [1.1 to 3.4] | 1.8 [1.7 to 1.9]

13. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from date of start of treatment to date of death due to any cause. If a patient was not known to have died, survival was censored at the date of last known date patient alive.
  OS was estimated using Kaplan-Meier estimates.
Time Frame: From start of treatment until death due to any cause, assessed up to 2 years for sabatolimab and 5.3 years for sabatolimab in combination with spartalizumab
Population: as for outcome 8
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 14 | 9 | 16 | 5 | 2 | 4 | 6 | 2 | 8 | 9 | 6 | 6 | 6 | 13 | 6 | 5 | 5 | 6 | 6 | 3 | 12 | 5 | 7 | 6 | 6 | 14 | 17 | 15 | 17 | 16
months | 4.1 [2.4 to 7.7] | 6.7 [4.6 to 9.2] | 10.3 [4.9 to 15.9] | 4.3 [1.4 to NA] — Not estimable due to insufficient number of participants with events. | 4.1 [1.8 to NA] — Not estimable due to insufficient number of participants with events. | 4.2 [2.3 to NA] — Not estimable due to insufficient number of participants with events. | 5.0 [1.7 to 7.5] | 8.5 [3.1 to NA] — Not estimable due to insufficient number of participants with events. | 12.5 [1.8 to NA] — Not estimable due to insufficient number of participants with events. | 2.5 [1.6 to 11.1] | 4.8 [2.8 to NA] — Not estimable due to insufficient number of participants with events. | 6.6 [1.9 to 11.5] | 24.4 [3.4 to NA] — Not estimable due to insufficient number of participants with events. | 10.0 [6.2 to 41.8] | 9.6 [1.5 to NA] — Not estimable due to insufficient number of participants with events. | 3.1 [1.2 to NA] — Not estimable due to insufficient number of participants with events. | 20.6 [2.0 to NA] — Not estimable due to insufficient number of participants with events. | 5.4 [0.5 to NA] — Not estimable due to insufficient number of participants with events. | NA [8.1 to NA] — Not estimable due to insufficient number of participants with events. | 3.6 [2.4 to NA] — Not estimable due to insufficient number of participants with events. | 8.6 [4.9 to 18.3] | 12.3 [3.7 to NA] — Not estimable due to insufficient number of participants with events. | 24.8 [1.5 to NA] — Not estimable due to insufficient number of participants with events. | 18.0 [1.4 to NA] — Not estimable due to insufficient number of participants with events. | 2.4 [0.2 to 6.8] | 4.0 [1.8 to 13.8] | 4.9 [3.4 to 11.2] | 10.9 [2.2 to 14.6] | 6.6 [1.1 to 9.0] | 6.7 [5.2 to 13.3]

14. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Sabatolimab
Description: Pharmacokinetic (PK) parameters were calculated based on sabatolimab serum concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed serum concentration following a dose.
Time Frame: pre-infusion and 1, 24, 168, 240 and 336 hours after completion of the sabatolimab infusion on Cycle 1 Day 1 and Cycle 3 Day 1. The duration of the infusion was 30 minutes. The duration of one cycle was 28 days.
Population: Patients in the pharmacokinetic analysis set (PAS) with an available value for the outcome measure in each timepoint. PAS consists of all patients who have at least one blood sample providing evaluable PK data.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 14 | 9 | 16 | 5 | 2 | 4 | 6 | 2 | 8 | 9 | 6 | 6 | 6 | 13 | 6 | 4 | 4 | 6 | 6 | 3 | 12 | 5 | 6 | 6 | 5 | 14 | 17 | 15 | 17 | 16
µg/mL
  Cycle 1 | 23 (6.28) | 81.3 (24.4) | 251 (57.3) | 429 (152) | 36.1 (0.919) | 74 (8.59) | 321 (64.2) | 443 (4.24) | 98.8 (50.8) | 271 (78.5) | 304 (86.5) | 457 (135) | 7.68 (3.68) | 23 (6.38) | 83 (20.7) | 58.3 (12.7) | 213 (4.19) | 189 (70.6) | 22.9 (5.91) | 23.3 (0.529) | 72 (18.3) | 59.7 (30.2) | 79 (26) | 254 (38.7) | 343 (112) | 34.6 (21.8) | 86.2 (27) | 394 (86.7) | 185 (64.6) | 233 (60.3)
  Cycle 3: number analyzed (Participants) | 8 | 5 | 10 | 1 | 0 | 0 | 3 | 1 | 2 | 2 | 1 | 2 | 6 | 8 | 3 | 1 | 3 | 2 | 4 | 2 | 8 | 4 | 5 | 4 | 1 | 6 | 5 | 4 | 8 | 9
  Cycle 3 | 24.8 (13.5) | 144 (60.8) | 420 (138) | 563 |  |  | 443 (190) | 709 | 116 (28.6) | 333 (39.6) | 448 | 713 (14.8) | 12.7 (16.8) | 40.2 (31.1) | 101 (25.6) | 45.4 | 379 (104) | 422 (49.5) | 25.8 (5.22) | 18.6 (0.99) | 77 (27.2) | 104 (32.5) | 102 (32.5) | 286 (60.8) | 557 | 31.2 (5.58) | 94.4 (19.1) | 412 (124) | 267 (82.5) | 316 (105)

15. Secondary Outcome: Time to Reach Maximum Serum Concentration (Tmax) of Sabatolimab
Description: PK parameters were calculated based on sabatolimab serum concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) serum concentration following a dose. Actual recorded sampling times were considered for the calculations.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Median (Full Range); unit: hours
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 14 | 9 | 16 | 5 | 2 | 4 | 6 | 2 | 8 | 9 | 6 | 6 | 6 | 13 | 6 | 4 | 4 | 6 | 6 | 3 | 12 | 5 | 6 | 6 | 4 | 14 | 17 | 15 | 15 | 16
hours
  Cycle 1 | 1.53 [1.5 to 2.08] | 1.5 [0.667 to 24.4] | 1.57 [1.42 to 1.88] | 1.53 [1.5 to 22.6] | 1.57 [1.53 to 1.6] | 1.57 [1.55 to 1.67] | 1.56 [1.5 to 1.62] | 1.53 [1.52 to 1.55] | 1.58 [1.5 to 2] | 1.5 [1.42 to 2.17] | 1.53 [1.48 to 23.2] | 1.55 [1.52 to 1.6] | 4 [4 to 4] | 3.08 [2.72 to 4.08] | 3.13 [1.53 to 4.08] | 3.09 [1.17 to 3.33] | 3.08 [1.6 to 3.47] | 3.48 [3.08 to 162] | 3.32 [3.08 to 3.55] | 3 [1.68 to 3.38] | 3.17 [2.52 to 4.12] | 3.25 [1.55 to 359] | 3.21 [3.07 to 21.9] | 3.08 [3 to 4] | 3.23 [3.05 to 26.3] | 1.5 [1.5 to 24.5] | 1.58 [1.5 to 140] | 1.67 [1.33 to 24.3] | 3.37 [3 to 164] | 3.15 [3 to 26]
  Cycle 3: number analyzed (Participants) | 8 | 5 | 10 | 1 | 0 | 0 | 3 | 1 | 2 | 2 | 1 | 2 | 1 | 8 | 3 | 0 | 3 | 2 | 3 | 1 | 8 | 4 | 5 | 4 | 1 | 6 | 5 | 4 | 8 | 6
  Cycle 3 | 1.54 [1.5 to 1.67] | 1.58 [0.583 to 24.5] | 1.53 [0.483 to 1.93] | 1.7 [1.7 to 1.7] |  |  | 1.55 [1.48 to 1.58] | 1.62 [1.62 to 1.62] | 1.21 [0.833 to 1.58] | 1.63 [1.58 to 1.67] | 1.5 [1.5 to 1.5] | 1.57 [1.55 to 1.58] | 3.25 [3.25 to 3.25] | 3.31 [3 to 164] | 3 [1.62 to 3.08] |  | 3.2 [3.03 to 3.3] | 3.04 [3 to 3.08] | 3.38 [3 to 19.7] | 3 [3 to 3] | 3.13 [2.9 to 24] | 3.04 [0 to 3.57] | 3.08 [3.08 to 3.23] | 3 [3 to 3.07] | 3.5 [3.5 to 3.5] | 1.58 [1.5 to 1.65] | 1.58 [1.5 to 1.7] | 1.58 [1.57 to 23.8] | 3.08 [1.43 to 25] | 3.24 [3.08 to 3.4]

16. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Sabatolimab
Description: PK parameters were calculated based on sabatolimab serum concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUClast calculation.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: day*µg/mL
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 14 | 9 | 16 | 5 | 2 | 4 | 6 | 2 | 7 | 8 | 6 | 6 | 1 | 12 | 6 | 4 | 4 | 5 | 6 | 3 | 12 | 5 | 6 | 6 | 4 | 12 | 17 | 15 | 15 | 16
day*µg/mL
  Cycle 1 | 128 (33.2) | 555 (191) | 1670 (438) | 2780 (862) | 231 (4.77) | 463 (47.9) | 2070 (570) | 3220 (107) | 851 (425) | 2290 (793) | 2800 (921) | 4480 (1610) | 86.5 | 126 (34.7) | 502 (146) | 393 (197) | 1550 (115) | 1450 (546) | 149 (63.1) | 109 (57.5) | 673 (245) | 606 (302) | 702 (329) | 1870 (570) | 3450 (2020) | 216 (85.3) | 805 (278) | 3710 (1280) | 1820 (735) | 2430 (988)
  Cycle 3: number analyzed (Participants) | 7 | 5 | 10 | 1 | 0 | 0 | 2 | 0 | 2 | 2 | 1 | 2 | 1 | 8 | 3 | 0 | 3 | 2 | 3 | 1 | 8 | 4 | 5 | 4 | 1 | 6 | 5 | 4 | 8 | 6
  Cycle 3 | 172 (157) | 1350 (576) | 3270 (900) | 4980 |  |  | 2300 (407) |  | 1100 (559) | 3590 (1120) | 2800 | 9080 (648) | 321 | 357 (356) | 824 (149) |  | 3110 (721) | 4040 (894) | 165 (57.3) | 124 | 710 (337) | 1310 (603) | 989 (425) | 2690 (1060) | 3530 | 223 (75.5) | 892 (499) | 3730 (1640) | 3060 (1230) | 4390 (1610)

17. Secondary Outcome: Terminal Elimination Half-life (T1/2) of Sabatolimab
Description: PK parameters were calculated based on sabatolimab serum concentrations by using non-compartmental methods. T1/2 was calculated by regression analysis of the terminal elimination phase. T1/2 was computed as 0.693/terminal elimination rate constant.
Time Frame: pre-infusion and 1, 24, 168, 240 and 336 hours after completion of the sabatolimab infusion on Cycle 3 Day 1. The duration of the infusion was 30 minutes. The duration of one cycle was 28 days.
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 5 | 3 | 9 | 1 | 0 | 0 | 2 | 0 | 2 | 2 | 1 | 2 | 1 | 7 | 2 | 0 | 3 | 2 | 3 | 1 | 8 | 4 | 5 | 4 | 1 | 5 | 5 | 3 | 7 | 6
days | 8.6 (4.9) | 16.5 (6.61) | 13.5 (5.1) | 33.8 |  |  | 12.1 (2.35) |  | 23.3 (11.1) | 13.7 (1.8) | 6.38 | 14.3 (13) | 17.5 | 13.7 (11.6) | 16.5 (7.69) |  | 17.6 (0.142) | 14.9 (6.72) | 6.46 (1.55) | 6.8 | 11.2 (5.27) | 16.4 (7.48) | 11.6 (3.66) | 13.9 (1.48) | 11.5 | 5.85 (1.77) | 12 (4.33) | 12.9 (5.62) | 19.1 (8.69) | 21.7 (2.14)

18. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Spartalizumab
Description: PK parameters were calculated based on spartalizumab serum concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed serum concentration following a dose.
Time Frame: pre-infusion and 1, 24, 168, 240 and 336 hours after completion of the spartalizumab infusion on Cycle 1 Day 1 and Cycle 3 Day 1. The duration of the infusion was 30 minutes. The duration of one cycle was 28 days.
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 6 | 13 | 6 | 4 | 5 | 6 | 6 | 3 | 12 | 5 | 7 | 6 | 6 | 17 | 16
µg/mL
  Cycle 1 | 21.3 (14.9) | 24.8 (7.8) | 20.1 (5.36) | 66.2 (12.2) | 18.6 (4.5) | 71.9 (23.8) | 28.8 (18.6) | 78.1 (35.2) | 24.3 (20.6) | 65.1 (23.1) | 121 (30) | 113 (27) | 112 (35.8) | 98.1 (29.1) | 126 (42.1)
  Cycle 3: number analyzed (Participants) | 6 | 8 | 3 | 1 | 3 | 2 | 4 | 2 | 8 | 4 | 5 | 4 | 1 | 8 | 9
  Cycle 3 | 38.4 (12) | 40.6 (7.09) | 34.5 (6.59) | 50 | 40.2 (6.12) | 125 (5.66) | 27 (3.77) | 122 (7.07) | 24 (12.5) | 97 (27.7) | 152 (40.2) | 134 (38.2) | 80.5 | 143 (46.5) | 174 (63.5)

19. Secondary Outcome: Time to Reach Maximum Serum Concentration (Tmax) of Spartalizumab
Description: PK parameters were calculated based on spartalizumab serum concentrations by using non-compartmental methods. Tmax is defined as the time to reach maximum (peak) serum concentration following a dose. Actual recorded sampling times were considered for the calculations.
Time Frame: as for outcome 18
Population: as for outcome 14
Measure: Median (Full Range); unit: hours
Arm/Group | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 6 | 12 | 6 | 4 | 5 | 5 | 6 | 3 | 12 | 5 | 7 | 6 | 5 | 15 | 16
hours
  Cycle 1 | 1.67 [1.52 to 23.3] | 1.58 [1.33 to 23.6] | 1.83 [1.5 to 23] | 1.63 [1.52 to 2.08] | 1.57 [1.5 to 23.3] | 1.67 [1.57 to 1.92] | 1.61 [1.52 to 1.75] | 1.58 [1.5 to 23.2] | 1.63 [1.1 to 22.2] | 1.53 [1.45 to 21.9] | 1.65 [1.57 to 22.6] | 1.5 [1.43 to 2] | 1.58 [1.55 to 1.68] | 1.58 [1.5 to 3] | 1.58 [1.37 to 2]
  Cycle 3: number analyzed (Participants) | 5 | 8 | 3 | 0 | 3 | 2 | 3 | 1 | 8 | 4 | 5 | 4 | 1 | 8 | 6
  Cycle 3 | 1.78 [1.53 to 21.2] | 1.5 [1.5 to 335] | 1.58 [1.5 to 21.2] |  | 1.58 [1.53 to 1.6] | 13 [1.5 to 24.6] | 1.72 [1.18 to 21.2] | 1.5 [1.5 to 1.5] | 1.5 [1.42 to 1.8] | 1.52 [1.5 to 1.58] | 1.58 [1.57 to 1.58] | 1.5 [1.5 to 1.57] | 165 [165 to 165] | 1.58 [1.5 to 24.5] | 1.56 [1.52 to 1.62]

20. Secondary Outcome: Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Spartalizumab
Description: PK parameters were calculated based on spartalizumab serum concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUClast calculation.
Time Frame: as for outcome 18
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: day*µg/mL
Arm/Group | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 5 | 12 | 6 | 4 | 5 | 5 | 6 | 3 | 12 | 5 | 7 | 6 | 5 | 15 | 16
day*µg/mL
  Cycle 1: number analyzed (Participants) | 4 | 12 | 6 | 4 | 5 | 5 | 6 | 3 | 12 | 5 | 7 | 6 | 5 | 15 | 16
  Cycle 1 | 197 (61.5) | 166 (44.3) | 160 (45.5) | 470 (173) | 152 (45.3) | 502 (157) | 279 (89.5) | 888 (452) | 291 (313) | 773 (289) | 1300 (735) | 1120 (366) | 1180 (501) | 1070 (322) | 1570 (747)
  Cycle 3: number analyzed (Participants) | 5 | 8 | 3 | 0 | 3 | 2 | 3 | 1 | 8 | 4 | 5 | 4 | 1 | 8 | 6
  Cycle 3 | 366 (147) | 389 (123) | 314 (43) |  | 348 (74.2) | 1280 (213) | 355 (58.4) | 1800 | 266 (154) | 1540 (558) | 2080 (837) | 1680 (610) | 1620 | 1870 (775) | 2890 (741)

21. Secondary Outcome: Terminal Elimination Half-life (T1/2) of Spartalizumab
Description: PK parameters were calculated based on spartalizumab serum concentrations by using non-compartmental methods. T1/2 was calculated by regression analysis of the terminal elimination phase. T1/2 was computed as 0.693/terminal elimination rate constant.
Time Frame: pre-infusion and 1, 24, 168, 240 and 336 hours after completion of the spartalizumab infusion on Cycle 3 Day 1. The duration of the infusion was 30 minutes. The duration of one cycle was 28 days.
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 4 | 7 | 2 | 0 | 2 | 2 | 3 | 1 | 8 | 3 | 5 | 4 | 1 | 7 | 5
days | 13.7 (6.46) | 19.9 (13.9) | 29.5 (19.4) |  | 13.2 (1.14) | 17.4 (9.53) | 30.6 (23.5) | 32.1 | 15.7 (5.6) | 23.6 (8.82) | 24.3 (9.72) | 22.9 (6.19) | 28.7 | 24.5 (11.8) | 22.7 (3.15)

22. Secondary Outcome: Number of Participants With Anti-sabatolimab Antibodies
Description: Immunogenicity was evaluated in serum in a validated three-tiered assay approach. Samples were screened for potential anti-sabatolimab antibodies and positive screen results were confirmed using a confirmatory assay. For confirmed anti-drug antibodies (ADA) positive samples, titers were determined. Patient ADA status was defined as follows:
  * ADA-negative at baseline: ADA-negative sample at baseline
  * ADA-positive at baseline: ADA-positive sample at baseline
  * ADA-negative post-baseline: patient with ADA-negative sample at baseline and at least 1 post baseline determinant sample, all of which are ADA-negative samples
  * ADA-inconclusive post-baseline = patient who does not qualify as ADA-positive or ADA-negative
  * Treatment-induced ADA-positive = ADA-negative sample at baseline and at least 1 treatment-induced ADA-positive sample
  * Treatment-boosted ADA-positive = ADA-positive sample at baseline and at least 1 treatment-boosted ADA-positive sample
Time Frame: Baseline (before first dose) and post-baseline (assessed throughout the treatment up to 1.9 years for sabatolimab and 4.9 years for sabatolimab in combination with spartalizumab)
Population: All patients who received at least one dose of assigned single agent sabatolimab, or at least one full or partial dose of assigned combination sabatolimab+spartalizumab and had a determinant baseline immunogenicity (IG) sample and at least one determinant post-baseline IG sample for assessing anti-sabatolimab antibodies. Determinant samples are defined as samples which are not unevaluable (where unevaluable = sample where assay is not available).
Measure: Number; unit: participants
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 8 | 8 | 14 | 5 | 2 | 4 | 6 | 2 | 5 | 7 | 5 | 6 | 6 | 13 | 5 | 5 | 4 | 5 | 6 | 2 | 12 | 5 | 5 | 6 | 2 | 11 | 13 | 12 | 13 | 14
participants
  ADA-negative at baseline: number analyzed (Participants) | 8 | 8 | 14 | 5 | 2 | 4 | 6 | 2 | 5 | 7 | 5 | 6 | 6 | 12 | 5 | 5 | 4 | 5 | 5 | 2 | 12 | 5 | 4 | 6 | 1 | 11 | 12 | 11 | 12 | 14
  ADA-negative at baseline | 5 | 8 | 14 | 5 | 2 | 4 | 6 | 2 | 5 | 7 | 5 | 6 | 6 | 12 | 4 | 5 | 4 | 4 | 5 | 2 | 12 | 5 | 4 | 5 | 1 | 9 | 12 | 10 | 11 | 13
  ADA-positive at baseline: number analyzed (Participants) | 8 | 8 | 14 | 5 | 2 | 4 | 6 | 2 | 5 | 7 | 5 | 6 | 6 | 12 | 5 | 5 | 4 | 5 | 5 | 2 | 12 | 5 | 4 | 6 | 1 | 11 | 12 | 11 | 12 | 14
  ADA-positive at baseline | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 1
  ADA-negative post-baseline: number analyzed (Participants) | 8 | 8 | 14 | 5 | 2 | 4 | 6 | 2 | 5 | 7 | 5 | 6 | 6 | 13 | 4 | 5 | 4 | 4 | 6 | 2 | 12 | 5 | 5 | 6 | 2 | 11 | 13 | 12 | 13 | 14
  ADA-negative post-baseline | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 5 | 5 | 0 | 2 | 0 | 0 | 3 | 1 | 10 | 0 | 1 | 0 | 0 | 8 | 5 | 2 | 1 | 0
  ADA- inconclusive post-baseline: number analyzed (Participants) | 8 | 8 | 14 | 5 | 2 | 4 | 6 | 2 | 5 | 7 | 5 | 6 | 6 | 13 | 4 | 5 | 4 | 4 | 6 | 2 | 12 | 5 | 5 | 6 | 2 | 11 | 13 | 12 | 13 | 14
  ADA- inconclusive post-baseline | 3 | 7 | 14 | 5 | 2 | 3 | 6 | 2 | 2 | 6 | 5 | 6 | 0 | 7 | 3 | 2 | 4 | 4 | 2 | 1 | 2 | 4 | 3 | 6 | 2 | 2 | 7 | 10 | 10 | 14
  Treatment-induced ADA-positive: number analyzed (Participants) | 8 | 8 | 14 | 5 | 2 | 4 | 6 | 2 | 5 | 7 | 5 | 6 | 6 | 13 | 4 | 5 | 4 | 4 | 6 | 2 | 12 | 5 | 5 | 6 | 2 | 11 | 13 | 12 | 13 | 14
  Treatment-induced ADA-positive | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0
  Treatment-boosted ADA-positive: number analyzed (Participants) | 8 | 8 | 14 | 5 | 2 | 4 | 6 | 2 | 5 | 7 | 5 | 6 | 6 | 13 | 4 | 5 | 4 | 4 | 6 | 2 | 12 | 5 | 5 | 6 | 2 | 11 | 13 | 12 | 13 | 14
  Treatment-boosted ADA-positive | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

23. Secondary Outcome: Number of Participants With Anti-spartalizumab Antibodies
Description: Immunogenicity was evaluated in serum in a validated three-tiered assay approach. Samples were screened for potential anti-spartalizumab antibodies and positive screen results were confirmed using a confirmatory assay. For confirmed anti-drug antibodies (ADA) positive samples, titers were determined. Patient ADA status was defined as follows:
  * ADA-negative at baseline: ADA-negative sample at baseline
  * ADA-positive at baseline: ADA-positive sample at baseline
  * ADA-negative post-baseline: patient with ADA-negative sample at baseline and at least 1 post baseline determinant sample, all of which are ADA-negative samples
  * ADA-inconclusive post-baseline = patient who does not qualify as ADA-positive or ADA-negative
  * Treatment-induced ADA-positive = ADA-negative sample at baseline and at least 1 treatment-induced ADA-positive sample
  * Treatment-boosted ADA-positive = ADA-positive sample at baseline and at least 1 treatment-boosted ADA-positive sample
Time Frame: Baseline (before first dose) and post-baseline (assessed throughout the treatment up to 4.9 years).
Population: All patients who received at least one full or partial dose of assigned combination sabatolimab+spartalizumab and had a determinant baseline immunogenicity (IG) sample and at least one determinant post-baseline IG sample for assessing anti-spartalizumab antibodies. Determinant samples are defined as samples which are not unevaluable (where unevaluable = sample where assay is not available).
Measure: Number; unit: participants
Arm/Group | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 5 | 12 | 5 | 5 | 4 | 5 | 6 | 2 | 11 | 5 | 4 | 6 | 3 | 13 | 13
participants
  ADA-negative at baseline: number analyzed (Participants) | 4 | 12 | 4 | 5 | 4 | 5 | 6 | 2 | 10 | 4 | 3 | 6 | 3 | 12 | 13
  ADA-negative at baseline | 4 | 9 | 3 | 5 | 4 | 4 | 5 | 2 | 9 | 4 | 3 | 6 | 3 | 12 | 13
  ADA-positive at baseline: number analyzed (Participants) | 4 | 12 | 4 | 5 | 4 | 5 | 6 | 2 | 10 | 4 | 3 | 6 | 3 | 12 | 13
  ADA-positive at baseline | 0 | 3 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  ADA-negative post-baseline: number analyzed (Participants) | 5 | 10 | 5 | 5 | 4 | 5 | 5 | 2 | 11 | 5 | 4 | 6 | 3 | 13 | 13
  ADA-negative post-baseline | 2 | 7 | 2 | 4 | 3 | 1 | 3 | 1 | 7 | 3 | 2 | 4 | 2 | 6 | 7
  ADA- inconclusive post-baseline: number analyzed (Participants) | 5 | 10 | 5 | 5 | 4 | 5 | 5 | 2 | 11 | 5 | 4 | 6 | 3 | 13 | 13
  ADA- inconclusive post-baseline | 1 | 1 | 2 | 1 | 1 | 4 | 1 | 1 | 2 | 2 | 2 | 1 | 1 | 6 | 6
  Treatment-induced ADA-positive: number analyzed (Participants) | 5 | 10 | 5 | 5 | 4 | 5 | 5 | 2 | 11 | 5 | 4 | 6 | 3 | 13 | 13
  Treatment-induced ADA-positive | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
  Treatment-boosted ADA-positive: number analyzed (Participants) | 5 | 10 | 5 | 5 | 4 | 5 | 5 | 2 | 11 | 5 | 4 | 6 | 3 | 13 | 13
  Treatment-boosted ADA-positive | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Baseline Expression of PD-L1
Description: The tumor expression of programmed cell death-ligand 1 (PD-L1) was measured by immunohistochemical methods. This record summarizes the baseline expression of PD-1 and the clinical benefit of study treatment. Clinical benefit (BOR: CR, PR, SD or NCRNPD) and No clinical benefit (BOR: PD) was based on local investigator assessment per RECIST v1.1.
Time Frame: Screening
Population: All patients who received at least one dose of assigned single agent sabatolimab, or at least one full or partial dose of assigned combination sabatolimab+spartalizumab and had a valid assessment for the outcome measure
Measure: Median (Full Range); unit: PD-L1 positivity percentage
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 8 | 5 | 9 | 5 | 2 | 4 | 5 | 2 | 4 | 3 | 3 | 6 | 5 | 9 | 4 | 4 | 4 | 3 | 4 | 1 | 11 | 3 | 4 | 6 | 3 | 11 | 14 | 11 | 10 | 14
PD-L1 positivity percentage
  Clinical benefit: number analyzed (Participants) | 2 | 2 | 4 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 3 | 4 | 6 | 1 | 0 | 1 | 1 | 2 | 0 | 4 | 2 | 3 | 3 | 0 | 4 | 2 | 4 | 5 | 2
  Clinical benefit | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 5.0] |  |  | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] |  | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] |  | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 10.0] | 1.25 [0.0 to 80.0] | 0.00 [0.0 to 0.0] |  | 5.00 [5.0 to 5.0] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] |  | 10.00 [0.0 to 90.0] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 1.0] | 0.00 [0.0 to 35.0] |  | 0.00 [0.0 to 0.5] | 22.50 [5.0 to 40.0] | 0.00 [0.0 to 1.0] | 80.0 [0.0 to 100.0] | 7.75 [0.5 to 15.0]
  No clinical benefit: number analyzed (Participants) | 6 | 3 | 5 | 5 | 2 | 3 | 4 | 2 | 3 | 2 | 3 | 3 | 1 | 3 | 3 | 4 | 3 | 2 | 2 | 1 | 7 | 1 | 1 | 3 | 3 | 7 | 12 | 7 | 5 | 12
  No clinical benefit | 0.00 [0.0 to 45.0] | 5.00 [0.0 to 80.0] | 0.00 [0.0 to 90.0] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] | 2.50 [0.0 to 5.0] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 90.0] | 0.00 [0.0 to 20.0] | 5.00 [5.0 to 5.0] | 0.50 [0.0 to 70.0] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 1.0] | 0.00 [0.0 to 0.0] | 2.50 [0.0 to 5.0] | 5.00 [0.0 to 10.0] | 40.00 [40.0 to 40.0] | 0.00 [0.0 to 80.0] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] | 0.00 [0.0 to 0.0] | 60.00 [5.0 to 70.0] | 0.00 [0.0 to 5.0] | 0.00 [0.0 to 1.0] | 0.00 [0.0 to 10.0] | 50.0 [0.0 to 100.0] | 1.00 [0.0 to 50.0]

25. Secondary Outcome: Baseline Expression of CD8+
Description: The tumor expression of CD8+ was measured by immunohistochemical methods. This record summarizes the baseline expression of CD8+ and the clinical benefit of study treatment. Clinical benefit (BOR: CR, PR, SD or NCRNPD) and No clinical benefit (BOR: PD) was based on local investigator assessment per RECIST v1.1.
Time Frame: Screening
Population: as for outcome 24
Measure: Median (Full Range); unit: percent marker area expression of CD8+
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 8 | 8 | 12 | 5 | 2 | 4 | 4 | 2 | 4 | 3 | 3 | 5 | 6 | 8 | 4 | 4 | 4 | 3 | 4 | 1 | 10 | 2 | 3 | 6 | 3 | 11 | 14 | 11 | 10 | 10
percent marker area expression of CD8+
  Clinical benefit: number analyzed (Participants) | 3 | 2 | 6 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 3 | 5 | 5 | 1 | 0 | 1 | 1 | 2 | 0 | 3 | 2 | 2 | 3 | 0 | 4 | 2 | 4 | 5 | 1
  Clinical benefit | 0.35 [0.1 to 2.0] | 0.35 [0.0 to 0.7] | 0.73 [0.3 to 35.8] |  |  | 1.00 [1.0 to 1.0] | 5.54 [5.54 to 5.54] |  | 0.04 [0.0 to 0.1] | 0.01 [0.01 to 0.01] |  | 0.26 [0.2 to 1.4] | 0.47 [0.2 to 3.6] | 2.07 [0.2 to 22.4] | 0.09 [0.09 to 0.09] |  | 8.32 [8.32 to 8.32] | 0.03 [0.03 to 0.03] | 0.08 [0.0 to 0.1] |  | 0.60 [0.0 to 54.0] | 3.81 [2.7 to 4.9] | 3.87 [0.1 to 7.7] | 0.55 [0.1 to 8.3] |  | 0.90 [0.3 to 1.3] | 0.60 [0.6 to 0.6] | 0.11 [0.0 to 0.6] | 7.08 [0.4 to 10.7] | 6.67 [6.67 to 6.67]
  No clinical benefit: number analyzed (Participants) | 5 | 6 | 6 | 5 | 2 | 3 | 3 | 2 | 2 | 2 | 3 | 2 | 1 | 3 | 3 | 4 | 3 | 2 | 2 | 1 | 7 | 0 | 1 | 3 | 3 | 7 | 12 | 7 | 5 | 9
  No clinical benefit | 2.17 [0.2 to 21.5] | 0.90 [0.2 to 1.4] | 0.13 [0.0 to 13.2] | 0.65 [0.5 to 0.7] | 4.28 [2.1 to 6.5] | 0.21 [0.0 to 4.3] | 0.37 [0.2 to 3.0] | 0.68 [0.0 to 1.3] | 0.29 [0.1 to 0.5] | 0.22 [0.1 to 0.3] | 0.55 [0.3 to 3.1] | 0.11 [0.11 to 0.11] | 4.76 [4.76 to 4.76] | 4.58 [3.6 to 6.2] | 1.25 [0.0 to 2.9] | 0.42 [0.0 to 7.7] | 0.16 [0.1 to 0.3] | 3.56 [2.9 to 4.3] | 0.10 [0.1 to 0.1] | 0.96 [0.96 to 0.96] | 0.59 [0.1 to 5.3] |  | 0.18 [0.18 to 0.18] | 0.12 [0.1 to 0.2] | 0.11 [0.1 to 0.2] | 0.16 [0.1 to 7.5] | 0.71 [0.1 to 4.2] | 0.38 [0.0 to 1.0] | 3.36 [0.8 to 4.5] | 3.47 [0.2 to 10.0]

26. Secondary Outcome: Baseline Expression of TIM-3
Description: The tumor expression of T-cell Immunoglobulin domain and Mucin domain-3 (TIM-3) was measured by immunohistochemical methods. This record summarizes the baseline expression of TIM-3 and the clinical benefit of study treatment. Clinical benefit (BOR: CR, PR, SD or NCRNPD) and No clinical benefit (BOR: PD) was based on local investigator assessment per RECIST v1.1.
Time Frame: Screening
Population: as for outcome 24
Measure: Median (Full Range); unit: percent marker area expression of TIM-3
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 8 | 5 | 9 | 4 | 2 | 3 | 5 | 2 | 2 | 3 | 3 | 6 | 5 | 8 | 4 | 4 | 3 | 3 | 4 | 1 | 10 | 3 | 4 | 6 | 2 | 11 | 14 | 11 | 9 | 10
percent marker area expression of TIM-3
  Clinical benefit: number analyzed (Participants) | 2 | 2 | 4 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3 | 4 | 5 | 1 | 0 | 0 | 1 | 2 | 0 | 3 | 2 | 3 | 3 | 0 | 4 | 2 | 4 | 4 | 1
  Clinical benefit | 3.01 [0.0 to 6.0] | 2.56 [2.56 to 2.6] | 6.68 [0.6 to 51.3] |  |  | 6.06 [6.06 to 6.06] | 41.00 [41.0 to 41.0] |  |  | 1.05 [1.05 to 1.05] |  | 6.26 [1.7 to 14.2] | 4.19 [0.3 to 6.5] | 15.19 [3.4 to 64.0] | 0.04 [0.04 to 0.04] |  |  | 0.66 [0.66 to 0.66] | 0.40 [0.2 to 0.6] |  | 7.13 [1.3 to 8.1] | 17.81 [8.9 to 26.8] | 11.27 [0.9 to 12.4] | 14.57 [0.7 to 20.3] |  | 5.05 [1.5 to 8.6] | 2.32 [0.9 to 3.7] | 1.66 [0.1 to 8.4] | 7.78 [2.5 to 21.8] | 28.92 [28.92 to 28.92]
  No clinical benefit: number analyzed (Participants) | 6 | 3 | 5 | 4 | 2 | 2 | 4 | 2 | 2 | 2 | 3 | 3 | 1 | 3 | 3 | 4 | 3 | 2 | 2 | 1 | 7 | 1 | 1 | 3 | 2 | 7 | 12 | 7 | 5 | 9
  No clinical benefit | 9.32 [0.1 to 49.2] | 6.10 [4.0 to 30.3] | 3.96 [1.2 to 28.9] | 0.99 [0.5 to 2.5] | 10.93 [7.2 to 14.7] | 0.88 [0.4 to 1.3] | 6.74 [1.3 to 10.9] | 5.49 [1.6 to 9.4] | 4.82 [0.7 to 8.9] | 2.70 [0.0 to 5.4] | 15.88 [1.4 to 20.7] | 2.36 [0.3 to 4.0] | 32.23 [32.23 to 32.23] | 47.27 [11.6 to 67.6] | 11.29 [0.5 to 30.1] | 7.27 [0.8 to 20.8] | 1.89 [0.3 to 11.3] | 8.92 [8.1 to 9.7] | 2.13 [0.2 to 4.1] | 52.24 [52.24 to 52.24] | 6.74 [3.5 to 17.2] | 0.84 [0.84 to 0.84] | 0.37 [0.37 to 0.37] | 2.88 [1.1 to 7.1] | 0.71 [0.6 to 0.8] | 1.50 [1.2 to 12.3] | 2.16 [0.1 to 22.9] | 6.20 [0.7 to 19.7] | 8.19 [6.7 to 28.0] | 3.11 [0.6 to 17.7]

27. Secondary Outcome: Baseline Expression of LAG-3
Description: The tumor expression of lymphocyte-activation gene-3 (LAG-3) was measured by immunohistochemical methods. This record summarizes the baseline expression of LAG-3 and the clinical benefit of study treatment. Clinical benefit (BOR: CR, PR, SD or NCRNPD) and No clinical benefit (BOR: PD) was based on local investigator assessment per RECIST v1.1.
Time Frame: Screening
Population: as for outcome 24
Measure: Median (Full Range); unit: percent marker area expression of LAG-3
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 8 | 4 | 8 | 4 | 2 | 3 | 4 | 2 | 3 | 2 | 3 | 6 | 5 | 8 | 4 | 4 | 3 | 3 | 4 | 1 | 10 | 2 | 4 | 6 | 3 | 11 | 12 | 11 | 10 | 12
percent marker area expression of LAG-3
  Clinical benefit: number analyzed (Participants) | 2 | 1 | 4 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 3 | 4 | 5 | 1 | 0 | 0 | 1 | 2 | 0 | 3 | 1 | 3 | 3 | 0 | 4 | 2 | 4 | 5 | 1
  Clinical benefit | 0.24 [0.0 to 0.5] | 0.08 [0.08 to 0.8] | 0.23 [0.0 to 26.2] |  |  | 1.30 [1.3 to 1.3] | 7.12 [7.12 to 7.12] |  | 0.03 [0.03 to 0.03] |  |  | 0.02 [0.0 to 0.3] | 0.31 [0.3 to 0.4] | 2.44 [0.0 to 32.1] | 0.00 [0.0 to 0.0] |  |  | 0.01 [0.01 to 0.01] | 0.01 [0.0 to 0.01] |  | 0.20 [0.1 to 0.2] | 2.08 [2.08 to 2.08] | 0.31 [0.0 to 1.7] | 0.83 [0.0 to 4.2] |  | 0.35 [0.1 to 1.1] | 0.16 [0.1 to 0.3] | 0.04 [0.0 to 0.5] | 3.08 [0.2 to 19.0] | 3.39 [3.39 to 3.39]
  No clinical benefit: number analyzed (Participants) | 6 | 3 | 4 | 4 | 2 | 2 | 3 | 2 | 2 | 2 | 3 | 3 | 1 | 3 | 3 | 4 | 3 | 2 | 2 | 1 | 7 | 1 | 1 | 3 | 3 | 7 | 10 | 7 | 5 | 11
  No clinical benefit | 1.61 [0.1 to 21.0] | 0.69 [0.4 to 4.8] | 2.68 [0.0 to 29.5] | 0.11 [0.0 to 0.3] | 2.11 [1.0 to 3.2] | 0.02 [0.01 to 0.02] | 0.14 [0.0 to 1.5] | 0.58 [0.0 to 1.2] | 0.10 [0.0 to 0.2] | 0.05 [0.0 to 0.1] | 0.18 [0.18 to 2.4] | 0.06 [0.0 to 0.1] | 7.63 [7.63 to 7.63] | 1.49 [0.9 to 6.2] | 0.78 [0.0 to 1.8] | 0.30 [0.1 to 2.4] | 0.05 [0.0 to 0.2] | 1.33 [1.1 to 1.6] | 0.07 [0.0 to 0.1] | 0.08 [0.08 to 0.08] | 0.33 [0.0 to 4.7] | 0.00 [0.0 to 0.0] | 0.05 [0.05 to 0.05] | 0.06 [0.0 to 0.1] | 0.03 [0.0 to 0.1] | 0.04 [0.0 to 4.0] | 0.43 [0.0 to 1.3] | 0.06 [0.0 to 0.8] | 1.98 [0.4 to 2.5] | 0.57 [0.0 to 10.0]

28. Secondary Outcome: Baseline Expression of CD163
Description: The tumor expression of CD163 was measured by immunohistochemical methods. This record summarizes the baseline expression of CD163 and the clinical benefit of study treatment. Clinical benefit (BOR: CR, PR, SD or NCRNPD) and No clinical benefit (BOR: PD) was based on local investigator assessment per RECIST v1.1.
Time Frame: Screening
Population: as for outcome 24
Measure: Median (Full Range); unit: percent marker area expression of CD163
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 8 | 8 | 13 | 5 | 2 | 3 | 4 | 2 | 4 | 3 | 3 | 6 | 6 | 8 | 4 | 4 | 4 | 3 | 4 | 1 | 10 | 2 | 3 | 6 | 3 | 10 | 12 | 11 | 8 | 10
percent marker area expression of CD163
  Clinical benefit: number analyzed (Participants) | 3 | 2 | 6 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 3 | 5 | 5 | 1 | 0 | 1 | 1 | 2 | 0 | 3 | 1 | 2 | 3 | 0 | 4 | 2 | 4 | 4 | 1
  Clinical benefit | 3.12 [1.0 to 20.5] | 0.26 [0.2 to 0.3] | 6.05 [0.5 to 40.2] |  |  | 14.56 [14.56 to 14.56] | 15.47 [15.47 to 15.47] |  | 0.42 [0.3 to 0.6] | 3.79 [3.79 to 3.79] |  | 5.53 [5.4 to 14.0] | 6.76 [1.8 to 10.2] | 21.36 [3.1 to 58.7] | 0.41 [0.41 to 0.41] |  | 12.93 [12.93 to 12.93] | 1.66 [1.66 to 1.66] | 3.44 [2.7 to 4.2] |  | 7.09 [4.2 to 8.9] | 26.40 [26.40 to 26.40] | 12.40 [4.2 to 20.6] | 5.46 [1.5 to 35.8] |  | 5.66 [4.4 to 7.7] | 7.41 [1.8 to 13.1] | 5.41 [0.1 to 13.1] | 16.34 [14.3 to 26.2] | 36.59 [36.59 to 36.59]
  No clinical benefit: number analyzed (Participants) | 5 | 6 | 7 | 5 | 2 | 2 | 3 | 2 | 2 | 2 | 3 | 3 | 1 | 3 | 3 | 4 | 3 | 2 | 2 | 1 | 7 | 1 | 1 | 3 | 3 | 6 | 10 | 7 | 4 | 9
  No clinical benefit | 11.53 [4.3 to 36.6] | 9.48 [3.4 to 14.8] | 5.22 [3.2 to 31.3] | 3.92 [0.8 to 4.9] | 7.60 [6.0 to 9.2] | 0.98 [0.9 to 1.0] | 14.30 [7.5 to 15.1] | 3.66 [2.2 to 5.1] | 6.95 [1.6 to 12.3] | 7.36 [1.7 to 13.0] | 19.69 [10.8 to 20.5] | 5.78 [1.9 to 7.7] | 16.17 [16.17 to 16.17] | 26.28 [24.3 to 70.4] | 6.23 [3.3 to 28.2] | 10.36 [4.6 to 289] | 5.08 [1.4 to 33.6] | 11.11 [4.7 to 17.5] | 1.14 [0.6 to 1.7] | 28.64 [28.64 to 28.64] | 10.62 [5.4 to 17.5] | 3.67 [3.67 to 3.67] | 1.41 [1.41 to 1.41] | 3.47 [2.5 to 23.1] | 5.80 [3.9 to 6.1] | 5.78 [0.6 to 18.5] | 4.92 [1.6 to 31.2] | 3.56 [2.0 to 11.6] | 17.46 [10.9 to 26.7] | 11.88 [4.0 to 54.8]

29. Secondary Outcome: Percentage Change From Baseline of Tumor Infiltrating Lymphocytes (TILs) Count
Description: The count of TILs was performed by hematoxylin and eosin stain.
Time Frame: Baseline (screening) and post-baseline (assessed throughout the treatment up to maximum 193 days)
Population: All patients who received at least one dose of assigned single agent sabatolimab, or at least one full or partial dose of assigned combination sabatolimab+spartalizumab and had a paired assessment at baseline and post-baseline for the outcome measure
Measure: Median (Full Range); unit: percentage change from baseline
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 2 | 2 | 6 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 2 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 2 | 1
percentage change from baseline | 41.67 [-50.0 to 133.3] | -100.00 [-100.0 to -100.0] | -25.00 [-100.0 to 900.0] |  | -50.00 [-50.0 to -50.0] |  |  |  |  |  |  | -70.00 [-100.0 to -40.0] | -75.00 [-100.0 to -50.0] | -66.67 [-66.67 to -66.67] | -25.00 [-50.0 to 0.0] | -50.00 [-50.0 to -50.0] | -50.00 [-100.0 to 0.0] |  |  | -97.50 [-97.5 to -97.5] | -87.50 [-87.5 to -87.5] |  |  |  |  | -66.67 [-100.0 to 100.0] | 550.00 [200.0 to 900.0] |  | -40.95 [-70.1 to -11.8] | -48.43 [-48.43 to -48.43]

30. Secondary Outcome: Phase II: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) During the On-treatment Period
Description: Number of participants with AEs and SAEs, including changes from baseline in vital signs, electrocardiograms and laboratory results qualifying and reported as AEs.
  AE grades to characterize the severity of the AEs were based on the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. For CTCAE v4.03, Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = death related to AE.
  The on-treatment period is defined from the day of first administration of study treatment up to 30 days after the date of its last administration.
Time Frame: From first dose of study medication up to 30 days after last dose, with a maximum duration of 3 years
Population: All patients in Phase II who received at least one full or partial dose of the combination sabatolimab+spartalizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 17 | 16
Participants
  AEs | 16 | 15
  Treatment-related AEs | 6 | 9
  AEs with grade ≥ 3 | 10 | 6
  Treatment-related AEs with grade ≥ 3 | 2 | 0
  SAEs | 9 | 2
  Fatal SAEs | 1 | 0
  AEs leading to discontinuation | 2 | 1
  AEs leading to dose adjustment/interruption | 4 | 0
  AEs requiring additional therapy | 15 | 14

31. Secondary Outcome: Phase II: Number of Participants With Dose Reductions and Dose Interruptions of Sabatolimab
Description: as for outcome 3
Time Frame: From first dose of study medication up to last dose, with a maximum duration of 2.9 years
Population: All patients in Phase II who received at least one full or partial dose of the combination sabatolimab+spartalizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 17 | 16
Participants
  At least one dose reduction | 0 | 0
  At least one dose interruption | 3 | 0

32. Secondary Outcome: Phase II: Number of Participants With Dose Reductions and Dose Interruptions of Spartalizumab
Description: as for outcome 4
Time Frame: From first dose of study medication up to last dose, with a maximum duration of 2.9 years
Population: All patients in Phase II who received at least one full or partial dose of the combination sabatolimab+spartalizumab
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 17 | 16
Participants
  At least one dose reduction | 0 | 0
  At least one dose interruption | 3 | 0

33. Secondary Outcome: Phase II: Dose Intensity of Sabatolimab
Description: Dose intensity of sabatolimab was calculated as cumulative actual dose in milligrams divided by duration of exposure in days and then multiplied by 28 days.
Time Frame: From first dose of study medication up to last dose, with a maximum duration of 2.9 years
Population: All patients in Phase II who received at least one full or partial dose of the combination sabatolimab+spartalizumab
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 17 | 16
milligrams | 772.94 (62.826) | 800.00 (0.000)

34. Secondary Outcome: Phase II: Dose Intensity of Spartalizumab
Description: Dose intensity of spartalizumab was calculated as cumulative actual dose in milligrams divided by duration of exposure in days and then multiplied by 28 days.
Time Frame: From first dose of study medication up to last dose, with a maximum duration of 2.9 years
Population: All patients in Phase II who received at least one full or partial dose of the combination sabatolimab+spartalizumab
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 17 | 16
milligrams | 386.47 (31.413) | 400.00 (0.000)

35. Post Hoc Outcome: All-Collected Deaths
Description: On-treatment and post-treatment safety follow-up deaths were collected from first dose of study medication to 30 days after last dose (sabatolimab single agent) and to 150 days after last dose (sabatolimab+spartalizumab). Survival follow-up deaths were collected from 31 days (sabatolimab) and 151 days (sabatolimab+spartalizumab) after last dose until end of study. All deaths refer to the sum of on-treatment and post-treatment safety follow-up deaths plus survival follow-up deaths.
Time Frame: On-treatment and post-treatment safety follow-up deaths: up to 2 years for sabatolimab and 5.3 years for sabatolimab + spartalizumab. Survival follow-up deaths: up to 2 years for sabatolimab and 5.3 years for sabatolimab + spartalizumab
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma
Number analyzed (Participants) | 14 | 9 | 16 | 5 | 2 | 4 | 6 | 2 | 8 | 9 | 6 | 6 | 6 | 13 | 6 | 5 | 5 | 6 | 6 | 3 | 12 | 5 | 7 | 6 | 6 | 14 | 17 | 15 | 17 | 16
participants
  On-treatment and post-treatment safety follow-up deaths | 9 | 4 | 6 | 5 | 1 | 4 | 5 | 1 | 3 | 4 | 4 | 3 | 1 | 5 | 2 | 5 | 2 | 3 | 0 | 3 | 5 | 2 | 1 | 2 | 4 | 8 | 9 | 6 | 9 | 6
  Survival follow-up deaths: number analyzed (Participants) | 5 | 5 | 10 | 0 | 1 | 0 | 1 | 1 | 5 | 5 | 2 | 3 | 5 | 8 | 4 | 0 | 3 | 3 | 6 | 0 | 7 | 3 | 6 | 4 | 2 | 6 | 8 | 9 | 8 | 10
  Survival follow-up deaths | 3 | 4 | 7 |  | 1 |  | 1 | 1 | 3 | 3 | 1 | 3 | 2 | 4 | 3 |  | 2 | 2 | 2 |  | 6 | 2 | 3 | 2 | 1 | 4 | 3 | 7 | 8 | 7
  All deaths | 12 | 8 | 13 | 5 | 2 | 4 | 6 | 2 | 6 | 7 | 5 | 6 | 3 | 9 | 5 | 5 | 4 | 5 | 2 | 3 | 11 | 4 | 4 | 4 | 5 | 12 | 12 | 13 | 17 | 13

ADVERSE EVENTS:
Time Frame: On-treatment and post-treatment safety follow-up: from first dose of study treatment to 30 days after last dose (sabatolimab) and to 150 days after last dose (sabatolimab+spartalizumab), up to 2 years for single agent and 5.3 years (phase Ib)/3.3 years (phase II) for combination. Deaths in survival period: from 31 days (single agent) and 151 days (combination) after last dose until end of study, up to 2 years for single agent and 5.3 years (phase Ib)/3.3 years (phase II) for combination.
Description: Deaths in the survival follow-up are not considered Adverse Events (AEs). No AEs were collected in the survival period.
Groups:
- Phase I Dose Escalation: MBG453 80mg Q2W ROW: Sabatolimab 80 mg every 2 weeks (Q2W) in Phase I Dose Escalation Part in rest of the world (ROW) patients. Safety data up to 30 days after last dose
- Phase I Dose Escalation: MBG453 240mg Q2W ROW: Sabatolimab 240 mg Q2W in Phase I Dose Escalation Part in ROW patients. Safety data up to 30 days after last dose
- Phase I Dose Escalation: MBG453 800mg Q2W ROW: Sabatolimab 800 mg Q2W in Phase I Dose Escalation Part in ROW patients. Safety data up to 30 days after last dose
- Phase I Dose Escalation: MBG453 1200mg Q2W ROW: Sabatolimab 1200 mg Q2W in Phase I Dose Escalation Part in ROW patients. Safety data up to 30 days after last dose
- Phase I Dose Escalation: MBG453 80mg Q2W Japan: Sabatolimab 80 mg Q2W in Phase I Dose Escalation Part in Japanese patients. Safety data up to 30 days after last dose
- Phase I Dose Escalation: MBG453 240mg Q2W Japan: Sabatolimab 240 mg Q2W in Phase I Dose Escalation Part in Japanese patients. Safety data up to 30 days after last dose
- Phase I Dose Escalation: MBG453 800mg Q2W Japan: Sabatolimab 800 mg Q2W in Phase I Dose Escalation Part in Japanese patients. Safety data up to 30 days after last dose
- Phase I Dose Escalation: MBG453 1200mg Q2W Japan: Sabatolimab 1200 mg Q2W in Phase I Dose Escalation Part in Japanese patients. Safety data up to 30 days after last dose
- Phase I Dose Escalation: MBG453 240mg Q4W ROW: Sabatolimab 240 mg every 4 weeks (Q4W) in Phase I Dose Escalation Part in ROW patients. Safety data up to 30 days after last dose
- Phase I Dose Escalation: MBG453 800mg Q4W ROW: Sabatolimab 800 mg Q4W in Phase I Dose Escalation Part in ROW patients. Safety data up to 30 days after last dose
- Phase I Dose Escalation: MBG453 1200mg Q4W ROW: Sabatolimab 1200 mg Q4W in Phase I Dose Escalation Part in ROW patients. Safety data up to 30 days after last dose
- Phase I Dose Escalation: MBG453 1200mg Q4W Japan: Sabatolimab 1200 mg Q4W in Phase I Dose Escalation Part in Japanese patients. Safety data up to 30 days after last dose
- Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W: Sabatolimab 20 mg Q2W in combination with spartalizumab 80 mg Q2W in Phase Ib Dose Escalation Part. Safety data up to 150 days after last dose
- Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W: Sabatolimab 80 mg Q2W in combination with spartalizumab 80 mg Q2W in Phase Ib Dose Escalation Part. Safety data up to 150 days after last dose
- Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W: Sabatolimab 240 mg Q2W in combination with spartalizumab 80 mg Q2W in Phase Ib Dose Escalation Part. Safety data up to 150 days after last dose
- Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W: Sabatolimab 240 mg Q2W in combination with spartalizumab 240 mg Q2W in Phase Ib Dose Escalation Part. Safety data up to 150 days after last dose
- Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W: Sabatolimab 800 mg Q2W in combination with spartalizumab 80 mg Q2W in Phase Ib Dose Escalation Part. Safety data up to 150 days after last dose
- Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W: Sabatolimab 800 mg Q2W in combination with spartalizumab 240 mg Q2W in Phase Ib Dose Escalation Part. Safety data up to 150 days after last dose
- Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W: Sabatolimab 80 mg Q4W in combination with spartalizumab 80 mg Q4W in Phase Ib Dose Escalation Part. Safety data up to 150 days after last dose
- Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W: Sabatolimab 80 mg Q4W in combination with spartalizumab 400 mg Q4W in Phase Ib Dose Escalation Part. Safety data up to 150 days after last dose
- Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W: Sabatolimab 240 mg Q4W in combination with spartalizumab 80 mg Q4W in Phase Ib Dose Escalation Part. Safety data up to 150 days after last dose
- Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W: Sabatolimab 240 mg Q4W in combination with spartalizumab 240 mg Q4W in Phase Ib Dose Escalation Part. Safety data up to 150 days after last dose
- Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W: Sabatolimab 240 mg Q4W in combination with spartalizumab 400 mg Q4W in Phase Ib Dose Escalation Part. Safety data up to 150 days after last dose
- Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W: Sabatolimab 800 mg Q4W in combination with spartalizumab 400 mg Q4W in Phase Ib Dose Escalation Part. Safety data up to 150 days after last dose
- Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W: Sabatolimab 1200 mg Q4W in combination with spartalizumab 400 mg Q4W in Phase Ib Dose Escalation Part. Safety data up to 150 days after last dose
- Dose Ranging Part: MBG453 80mg Q4W: Sabatolimab 80 mg Q4W in Dose Ranging Part. Safety data up to 30 days after last dose
- Dose Ranging Part: MBG453 240mg Q4W: Sabatolimab 240 mg Q4W in Dose Ranging Part. Safety data up to 30 days after last dose
- Dose Ranging Part: MBG453 1200mg Q4W: Sabatolimab 1200 mg Q4W in Dose Ranging Part. Safety data up to 30 days after last dose
- Phase II: MBG453 + PDR001 NSCLC: Sabatolimab 800 mg Q4W in combination with spartalizumab 400 mg Q4W in non-small cell lung carcinoma (NSCLC). Safety data up to 150 days after last dose
- Phase II: MBG453 + PDR001 Melanoma: Sabatolimab 800 mg Q4W in combination with spartalizumab 400 mg Q4W in melanoma. Safety data up to 150 days after last dose
- Phase I Dose Escalation: MBG453 80mg Q2W ROW - Survival Period; Phase I Dose Escalation: MBG453 240mg Q2W ROW - Survival Period; Phase I Dose Escalation: MBG453 800mg Q2W ROW - Survival Period; Phase I Dose Escalation: MBG453 1200mg Q2W ROW - Survival Period; Phase I Dose Escalation: MBG453 80mg Q2W Japan - Survival Period; Phase I Dose Escalation: MBG453 240mg Q2W Japan - Survival Period; Phase I Dose Escalation: MBG453 800mg Q2W Japan - Survival Period; Phase I Dose Escalation: MBG453 1200mg Q2W Japan - Survival Period; Phase I Dose Escalation: MBG453 240mg Q4W ROW - Survival Period; Phase I Dose Escalation: MBG453 800mg Q4W ROW - Survival Period; Phase I Dose Escalation: MBG453 1200mg Q4W ROW - Survival Period; Phase I Dose Escalation: MBG453 1200mg Q4W Japan - Survival Period; Dose Ranging Part: MBG453 80mg Q4W - Survival Period; Dose Ranging Part: MBG453 240mg Q4W - Survival Period; Dose Ranging Part: MBG453 1200mg Q4W - Survival Period: Deaths collected in the survival follow-up period (starting from Day 31 post-treatment for sabatolimab single agent). No AEs were collected during this period.
- Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W - Survival Period; Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W - Survival Period; Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W - Survival Period; Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W - Survival Period; Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W - Survival Period; Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W - Survival Period; Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W - Survival Period; Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W - Survival Period; Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W - Survival Period; Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W - Survival Period; Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W - Survival Period; Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W - Survival Period; Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W - Survival Period; Phase II: MBG453 + PDR001 NSCLC - Survival Period; Phase II: MBG453 + PDR001 Melanoma - Survival Period: Deaths collected in the survival follow-up period (starting from Day 151 post-treatment for sabatolimab+spartalizumab). No AEs were collected during this period.
Arm/Group | Phase I Dose Escalation: MBG453 80mg Q2W ROW | Phase I Dose Escalation: MBG453 240mg Q2W ROW | Phase I Dose Escalation: MBG453 800mg Q2W ROW | Phase I Dose Escalation: MBG453 1200mg Q2W ROW | Phase I Dose Escalation: MBG453 80mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q2W Japan | Phase I Dose Escalation: MBG453 800mg Q2W Japan | Phase I Dose Escalation: MBG453 1200mg Q2W Japan | Phase I Dose Escalation: MBG453 240mg Q4W ROW | Phase I Dose Escalation: MBG453 800mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W ROW | Phase I Dose Escalation: MBG453 1200mg Q4W Japan | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W | Dose Ranging Part: MBG453 80mg Q4W | Dose Ranging Part: MBG453 240mg Q4W | Dose Ranging Part: MBG453 1200mg Q4W | Phase II: MBG453 + PDR001 NSCLC | Phase II: MBG453 + PDR001 Melanoma | Phase I Dose Escalation: MBG453 80mg Q2W ROW - Survival Period | Phase I Dose Escalation: MBG453 240mg Q2W ROW - Survival Period | Phase I Dose Escalation: MBG453 800mg Q2W ROW - Survival Period | Phase I Dose Escalation: MBG453 1200mg Q2W ROW - Survival Period | Phase I Dose Escalation: MBG453 80mg Q2W Japan - Survival Period | Phase I Dose Escalation: MBG453 240mg Q2W Japan - Survival Period | Phase I Dose Escalation: MBG453 800mg Q2W Japan - Survival Period | Phase I Dose Escalation: MBG453 1200mg Q2W Japan - Survival Period | Phase I Dose Escalation: MBG453 240mg Q4W ROW - Survival Period | Phase I Dose Escalation: MBG453 800mg Q4W ROW - Survival Period | Phase I Dose Escalation: MBG453 1200mg Q4W ROW - Survival Period | Phase I Dose Escalation: MBG453 1200mg Q4W Japan - Survival Period | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W - Survival Period | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W - Survival Period | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W - Survival Period | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W - Survival Period | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W - Survival Period | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W - Survival Period | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W - Survival Period | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W - Survival Period | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W - Survival Period | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W - Survival Period | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W - Survival Period | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W - Survival Period | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W - Survival Period | Dose Ranging Part: MBG453 80mg Q4W - Survival Period | Dose Ranging Part: MBG453 240mg Q4W - Survival Period | Dose Ranging Part: MBG453 1200mg Q4W - Survival Period | Phase II: MBG453 + PDR001 NSCLC - Survival Period | Phase II: MBG453 + PDR001 Melanoma - Survival Period
All-Cause Mortality (participants affected / at risk) | 9/14 | 4/9 | 6/16 | 5/5 | 1/2 | 4/4 | 5/6 | 1/2 | 3/8 | 4/9 | 4/6 | 3/6 | 1/6 | 5/13 | 2/6 | 5/5 | 2/5 | 3/6 | 0/6 | 3/3 | 5/12 | 2/5 | 1/7 | 2/6 | 4/6 | 8/14 | 9/17 | 6/15 | 9/17 | 6/16 | 3/5 | 4/5 | 7/10 | 0/0 | 1/1 | 0/0 | 1/1 | 1/1 | 3/5 | 3/5 | 1/2 | 3/3 | 2/5 | 4/8 | 3/4 | 0/0 | 2/3 | 2/3 | 2/6 | 0/0 | 6/7 | 2/3 | 3/6 | 2/4 | 1/2 | 4/6 | 3/8 | 7/9 | 8/8 | 7/10
Serious Adverse Events (participants affected / at risk) | 6/14 | 1/9 | 9/16 | 2/5 | 0/2 | 0/4 | 0/6 | 0/2 | 3/8 | 6/9 | 4/6 | 0/6 | 2/6 | 7/13 | 2/6 | 5/5 | 4/5 | 0/6 | 4/6 | 1/3 | 2/12 | 3/5 | 2/7 | 4/6 | 5/6 | 10/14 | 8/17 | 9/15 | 9/17 | 5/16 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 13/14 | 9/9 | 14/16 | 5/5 | 2/2 | 4/4 | 6/6 | 2/2 | 7/8 | 9/9 | 5/6 | 6/6 | 6/6 | 12/13 | 6/6 | 5/5 | 5/5 | 6/6 | 6/6 | 3/3 | 11/12 | 5/5 | 6/7 | 6/6 | 6/6 | 13/14 | 17/17 | 14/15 | 17/17 | 15/16 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Escalation: MBG453 80mg Q2W ROW (N=14) | Phase I Dose Escalation: MBG453 240mg Q2W ROW (N=9) | Phase I Dose Escalation: MBG453 800mg Q2W ROW (N=16) | Phase I Dose Escalation: MBG453 1200mg Q2W ROW (N=5) | Phase I Dose Escalation: MBG453 80mg Q2W Japan (N=2) | Phase I Dose Escalation: MBG453 240mg Q2W Japan (N=4) | Phase I Dose Escalation: MBG453 800mg Q2W Japan (N=6) | Phase I Dose Escalation: MBG453 1200mg Q2W Japan (N=2) | Phase I Dose Escalation: MBG453 240mg Q4W ROW (N=8) | Phase I Dose Escalation: MBG453 800mg Q4W ROW (N=9) | Phase I Dose Escalation: MBG453 1200mg Q4W ROW (N=6) | Phase I Dose Escalation: MBG453 1200mg Q4W Japan (N=6) | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W (N=6) | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W (N=13) | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W (N=6) | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W (N=5) | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W (N=5) | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W (N=6) | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W (N=6) | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W (N=3) | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W (N=12) | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W (N=5) | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W (N=7) | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W (N=6) | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W (N=6) | Dose Ranging Part: MBG453 80mg Q4W (N=14) | Dose Ranging Part: MBG453 240mg Q4W (N=17) | Dose Ranging Part: MBG453 1200mg Q4W (N=15) | Phase II: MBG453 + PDR001 NSCLC (N=17) | Phase II: MBG453 + PDR001 Melanoma (N=16) | Phase I Dose Escalation: MBG453 80mg Q2W ROW - Survival Period (N=0) | Phase I Dose Escalation: MBG453 240mg Q2W ROW - Survival Period (N=0) | Phase I Dose Escalation: MBG453 800mg Q2W ROW - Survival Period (N=0) | Phase I Dose Escalation: MBG453 1200mg Q2W ROW - Survival Period (N=0) | Phase I Dose Escalation: MBG453 80mg Q2W Japan - Survival Period (N=0) | Phase I Dose Escalation: MBG453 240mg Q2W Japan - Survival Period (N=0) | Phase I Dose Escalation: MBG453 800mg Q2W Japan - Survival Period (N=0) | Phase I Dose Escalation: MBG453 1200mg Q2W Japan - Survival Period (N=0) | Phase I Dose Escalation: MBG453 240mg Q4W ROW - Survival Period (N=0) | Phase I Dose Escalation: MBG453 800mg Q4W ROW - Survival Period (N=0) | Phase I Dose Escalation: MBG453 1200mg Q4W ROW - Survival Period (N=0) | Phase I Dose Escalation: MBG453 1200mg Q4W Japan - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W - Survival Period (N=0) | Dose Ranging Part: MBG453 80mg Q4W - Survival Period (N=0) | Dose Ranging Part: MBG453 240mg Q4W - Survival Period (N=0) | Dose Ranging Part: MBG453 1200mg Q4W - Survival Period (N=0) | Phase II: MBG453 + PDR001 NSCLC - Survival Period (N=0) | Phase II: MBG453 + PDR001 Melanoma - Survival Period (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Left ventricular dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Duodenal stenosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oesophageal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pyrexia (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Campylobacter gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Meningoencephalitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pleural infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Serratia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pericardial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Embolic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Mental disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Inferior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Escalation: MBG453 80mg Q2W ROW (N=14) | Phase I Dose Escalation: MBG453 240mg Q2W ROW (N=9) | Phase I Dose Escalation: MBG453 800mg Q2W ROW (N=16) | Phase I Dose Escalation: MBG453 1200mg Q2W ROW (N=5) | Phase I Dose Escalation: MBG453 80mg Q2W Japan (N=2) | Phase I Dose Escalation: MBG453 240mg Q2W Japan (N=4) | Phase I Dose Escalation: MBG453 800mg Q2W Japan (N=6) | Phase I Dose Escalation: MBG453 1200mg Q2W Japan (N=2) | Phase I Dose Escalation: MBG453 240mg Q4W ROW (N=8) | Phase I Dose Escalation: MBG453 800mg Q4W ROW (N=9) | Phase I Dose Escalation: MBG453 1200mg Q4W ROW (N=6) | Phase I Dose Escalation: MBG453 1200mg Q4W Japan (N=6) | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W (N=6) | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W (N=13) | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W (N=6) | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W (N=5) | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W (N=5) | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W (N=6) | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W (N=6) | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W (N=3) | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W (N=12) | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W (N=5) | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W (N=7) | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W (N=6) | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W (N=6) | Dose Ranging Part: MBG453 80mg Q4W (N=14) | Dose Ranging Part: MBG453 240mg Q4W (N=17) | Dose Ranging Part: MBG453 1200mg Q4W (N=15) | Phase II: MBG453 + PDR001 NSCLC (N=17) | Phase II: MBG453 + PDR001 Melanoma (N=16) | Phase I Dose Escalation: MBG453 80mg Q2W ROW - Survival Period (N=0) | Phase I Dose Escalation: MBG453 240mg Q2W ROW - Survival Period (N=0) | Phase I Dose Escalation: MBG453 800mg Q2W ROW - Survival Period (N=0) | Phase I Dose Escalation: MBG453 1200mg Q2W ROW - Survival Period (N=0) | Phase I Dose Escalation: MBG453 80mg Q2W Japan - Survival Period (N=0) | Phase I Dose Escalation: MBG453 240mg Q2W Japan - Survival Period (N=0) | Phase I Dose Escalation: MBG453 800mg Q2W Japan - Survival Period (N=0) | Phase I Dose Escalation: MBG453 1200mg Q2W Japan - Survival Period (N=0) | Phase I Dose Escalation: MBG453 240mg Q4W ROW - Survival Period (N=0) | Phase I Dose Escalation: MBG453 800mg Q4W ROW - Survival Period (N=0) | Phase I Dose Escalation: MBG453 1200mg Q4W ROW - Survival Period (N=0) | Phase I Dose Escalation: MBG453 1200mg Q4W Japan - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 20mg Q2W + PDR001 80mg Q2W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 80mg Q2W + PDR001 80mg Q2W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 80mg Q2W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 240mg Q2W + PDR001 240mg Q2W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 80mg Q2W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 800mg Q2W + PDR001 240mg Q2W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 80mg Q4W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 80mg Q4W + PDR001 400mg Q4W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 80mg Q4W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 240mg Q4W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 240mg Q4W + PDR001 400mg Q4W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 800mg Q4W + PDR001 400mg Q4W - Survival Period (N=0) | Phase Ib Dose Escalation: MBG453 1200mg Q4W + PDR001 400mg Q4W - Survival Period (N=0) | Dose Ranging Part: MBG453 80mg Q4W - Survival Period (N=0) | Dose Ranging Part: MBG453 240mg Q4W - Survival Period (N=0) | Dose Ranging Part: MBG453 1200mg Q4W - Survival Period (N=0) | Phase II: MBG453 + PDR001 NSCLC - Survival Period (N=0) | Phase II: MBG453 + PDR001 Melanoma - Survival Period (N=0)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 2 | 0 | 0 | 0 | 2 | 2 | 3 | 3 | 1 | 3 | 1 | 3 | 1 | 1 | 1 | 0 | 1 | 2 | 2 | 1 | 1 | 1 | 2 | 1 | 4 | 5 | 4 | 4 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Normocytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Atrial thrombosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hydrocele (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cushing's syndrome (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperprolactinaemia (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypopituitarism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Eye paraesthesia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Foreign body sensation in eyes (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lacrimation increased (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vitreous floaters (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 0 | 3 | 0 | 1 | 0 | 2 | 3 | 0 | 2 | 3 | 2 | 3 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal pain lower (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Ascites (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 2 | 3 | 2 | 1 | 1 | 0 | 1 | 1 | 4 | 0 | 1 | 0 | 1 | 3 | 2 | 0 | 1 | 0 | 3 | 1 | 4 | 0 | 1 | 1 | 0 | 4 | 4 | 2 | 5 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 2 | 3 | 4 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 2 | 2 | 0 | 1 | 1 | 2 | 3 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 3 | 1 | 3 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Large intestinal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 5 | 1 | 5 | 0 | 0 | 0 | 5 | 1 | 1 | 3 | 3 | 1 | 0 | 2 | 1 | 1 | 0 | 1 | 3 | 1 | 2 | 1 | 0 | 2 | 0 | 4 | 3 | 3 | 3 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oral discharge (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rectal tenesmus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 2 | 2 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 4 | 0 | 2 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Asthenia (General disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Axillary pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Chest discomfort (General disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Chills (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Early satiety (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Facial pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Fatigue (General disorders) | 4 | 5 | 6 | 2 | 0 | 0 | 4 | 0 | 2 | 2 | 1 | 2 | 1 | 7 | 3 | 2 | 2 | 0 | 2 | 1 | 3 | 3 | 1 | 1 | 1 | 4 | 4 | 6 | 3 | 5 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Generalised oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperpyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Malaise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Nodule (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oedema peripheral (General disorders) | 2 | 1 | 1 | 0 | 1 | 1 | 2 | 2 | 1 | 1 | 1 | 3 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pain (General disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pyrexia (General disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 3 | 1 | 0 | 1 | 2 | 2 | 0 | 1 | 0 | 1 | 4 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 4 | 4 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vascular device occlusion (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Xerosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Contrast media allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Aerococcus urinae infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dermatophytosis of nail (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gastrointestinal viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hepatitis B reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Infected cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Kidney infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lip infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lower respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oral fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Parotitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Streptococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Upper aerodigestive tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Viral rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Ammonia increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Amylase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Aspartate aminotransferase (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 2 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood creatine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood creatinine increased (Investigations) | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood potassium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Body temperature increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Coronavirus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Human chorionic gonadotropin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 2 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Low density lipoprotein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Platelet count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Weight decreased (Investigations) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 6 | 1 | 2 | 0 | 0 | 2 | 4 | 1 | 1 | 1 | 3 | 3 | 2 | 2 | 2 | 1 | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 2 | 0 | 1 | 4 | 2 | 1 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Folate deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 3 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypouricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypovitaminosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 4 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 3 | 2 | 2 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 1 | 2 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Fracture pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 2 | 4 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Aphasia (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Ataxia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Brain oedema (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cranial nerve disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Diabetic neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dizziness (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dizziness postural (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dysaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Facial paralysis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Facial paresis (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Headache (Nervous system disorders) | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypoglossal nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Migraine (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Muscle spasticity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Myasthenia gravis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Anxiety (Psychiatric disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Confusional state (Psychiatric disorders) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Bladder spasm (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Renal disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Strangury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pelvic discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vaginal odour (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vulvovaginal erythema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 4 | 3 | 1 | 0 | 3 | 0 | 1 | 0 | 3 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 3 | 3 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 4 | 1 | 0 | 1 | 2 | 0 | 3 | 1 | 2 | 1 | 0 | 3 | 0 | 1 | 3 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 1 | 2 | 3 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pulmonary artery aneurysm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 2 | 2 | 0 | 0 | 1 | 1 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 2 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Menopause (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypertension (Vascular disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Hypotension (Vascular disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Peripheral embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Subclavian vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA
Venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/68/NCT02608268/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-29): https://cdn.clinicaltrials.gov/large-docs/68/NCT02608268/SAP_001.pdf